**Official Title:** A multicenter, randomized, double-blind, placebo-controlled, phase 3 study to evaluate the efficacy and safety, of SA237 as monotherapy in

patients with neuromyelitis optica (NMO) and neuromyelitis optica

spectrum disorder (NMOSD)

NCT Number: NCT02073279

**Document Date:** SAP Version 7: 26-Nov-18



Chugai Pharmaceutical Co. Ltd.

**SA-309JG** 

A multicenter, randomized, double-blind, placebo-controlled, phase 3 study to evaluate the efficacy and safety, of SA237 as monotherapy in patients with neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD)

Statistical Analysis Plan

PAREXEL Project Number: 214545

Version 7.0

Date: 26NOV2018


# SIGNATURE PAGE

Approved by:

28 Nov 2018 Date


Related to: SOP-GDO-WW-019

# PAREXEL SIGNATURE PAGE

This document has been signed electronically on the final page by the following:

| Author | Signatory |
|--------|---------------|
| | Project Role: |

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018


# TABLE OF CONTENTS

| 1 | IN | TRODU | JCTION | | . 8 |
|---|---|---|---|---|---|
| 2 | ST | TUDY C | BJECTIVES | | . 8 |
| 3 | IN | VESTI | GATIONAL PI | LAN | . 8 |
| | 3.1 | Overal | Study Design | and Plan | . 8 |
| | 3.2 | Efficac | y and Safety V | ariables | . 9 |
| | 3.2. | 1 | Efficacy Varia | ables | . 9 |
| | 3.2. | 2 | Safety Variab | les | 10 |
| 4 | ST | TATIST: | CAL METHO | DDS | 10 |
| | 4.1 | Data Q | uality Assuran | ce | 10 |
| | 4.2 | Genera | l Presentation ( | Considerations | 10 |
| | 4.3 | Handli | ng of Missing o | dates | 12 |
| | 4.4 | Study S | Subjects | | 13 |
| | | 4.4.1 I | Disposition of S | Subjects | 13 |
| | | | | tions | |
| | | and the state of t | the second of th | | |
| | | | | seline Characteristics | |
| | | | | nt Medications | |
| | | | The second control of the second control of | e | |
| | 4.10 | | * | | |
| | | 4.10.1 | | Data Conventions | |
| | | | | ti-center Studies | |
| | | | · | istments for Covariates | |
| | | | | dling of Dropouts or Missing Data | |
| | | | | tiple Comparisons/Multiplicity | |
| | | | | mination of Subgroups | |
| | | | 20.00 | 5D Scoring Algorithm | |
| | | | | 36 Scoring Algorithm | |
| | | | | CIT-Fatigue Scale Scoring Algorithm | |
| | | | | SS Scoring | |
| | | | | RS Scoring | |
| | | | | BI Scoring | |
| | | | | isual acuity function (Snellen chart) | |
| | | | Water and the second of the second of the second | acy Variable | |
| | | 4.10.3 | | ficacy Variables | |
| | | | the second secon | Secondary Endpoints | |
| | grades | | | er Secondary Endpoints | |
| | 4.11 | The second second second second second | | Jenna | |
| | | | (1774) P. | llyses | |
| | | | SALES SALES CONTRACTOR AND AND AND ADDRESS OF THE SALES O | oosure | |
| | | T.11.J | Mayerse Evel | 11.3 | _C |

| | | 4.11.4 Deaths, Serious Adverse Events, and Other Significant Adverse Events | 29 |
|---|---|---|---|
| | | 4.11.5 C-SSRS | 29 |
| | | 4.11.6 Adverse event of special interest (AESI) | 29 |
| | | 4.11.5 Selected Adverse Events | |
| | | 4.11.7 Infections, Serious Infection, | 30 |
| | | 4.11.8 Anaphylaxis | 30 |
| | | 4.11.9 IRR and ISR | 31 |
| | | 4.11.10 Clinical Laboratory Evaluation | 31 |
| | | 4.11.11 AST and ALT: | 32 |
| | | 4.11.12 Electrocardiograms | |
| | | 4.11.13 Vital Signs, Physical Findings and Other Observations Related to Safety | 33 |
| | 4.12 | 2 Pharmacokinetics and Pharmacodynamics | 33 |
| | 4.13 | 3 Immunogenicity | 36 |
| | | Determination of Sample Size | |
| 5 | Cl | hanges in the Conduct of the Study or Planned Analysis | 40 |
| | 5.1 | Amendment from Ver 1.0 to 2.0 | 40 |
| | 5.2 | Amendment from Ver 2.0 to 3.0 | 40 |
| | 5.3 | Amendment from Ver 3.0 to 4.0 | 40 |
| | 5.4 | Amendment from Ver 4.0 to 5.0 | 40 |
| | 5.5 | Amendment from Ver 5.0 to 6.0 | 40 |
| | 5.6 | Amendment from Ver 6.0 to 6.1 | 41 |
| | 5.7 | Amendment from Ver 6.1 to 7.0 | 41 |
| 6 | RI | EFERENCES | 42 |
| 7 | A | PPENDIX | 43 |
| | 7.1 | SAS code for primary and key secondary analysis | 43 |
| | | EQ-5D Scoring Algorithm: | |
| | | Procedure to identify the clinical relapse of optic neuritis occurred in the double-blind | |
| | | period: 52 | |
| | | MedDRA basket | |
| | 7.5 | Laboratory Data Conversion and Transformation Rules | 56 |
| | 7.6 | Rule for summary of titer for anti AQP4 antibody status | 60 |

#### LIST OF ABBREVIATIONS

AE(s) Adverse event(s)

Analysis of covariance **ANCOVA** 

**ATC** Anatomical Therapeutic and Chemical

AQP4 Aquaporin-4

ARR Annualized relapse rate

Baseline observation carried forward **BOCF** 

**CEC** Clinical Endpoint Committee

C-SSRS Columbia-Suicide Severity Rating Scale

CV Coefficient of Variation

**eCRF** Electronic Case Report form

**ECG** Electrocardiogram

**EDSS Expanded Disability Status Scale** 

**FACIT** Functional Assessment Of Chronic Illness Therapy

**FPI** First patient in

Generalized Estimating Equation **GEE** 

ITT Intent-to-treat

LLOO Lower Limit of Quantification

MedDRA Medical Dictionary for Regulatory Activities

**MMRM** Mixed-effect model repeated measures

mRS Modified Rankin Scale **NMO** Neuromyelitis optica

**NMOSD** NMO spectrum disorder

Pharmacodynamics PD PK Pharmacokinetics

Pharmacokinetic Per-Protocol Set **PK-PPS** 

**PPS** Per-Protocol Set PT Preferred term Q4W Every 4 Weeks

Serious adverse event(s) SAE(s) SAP Statistical analysis plan

SC Subcutaneously

SD Standard deviation

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019

Short Form Generic Health Survey SF-36

SF-MPQ Short Form McGill Pain Questionnaire

**SFU** Safety Follow-Up

SOC System organ class

Safety Set SAF

Time to first relapse TFR Visual Analogue Scale VAS

World Health Organization Drug Dictionary WHO-DD

Zarit Burden Interview ZBI

TP-GDO-WW-016-01 Confidential Version 7.0 Version Date: 28NOV2018


#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) provides details of the summaries and analyses to be performed to report the results of the study. It should be read in conjunction with following documents:

- Study Protocol, Version 8.2AB, 25th October 2018
- Electronic Case Report Form (eCRF), Version 10.0, 22<sup>nd</sup> December 2017

#### 2 STUDY OBJECTIVES

The objective of this study is to evaluate the efficacy and safety of SA237 monotherapy in patients with neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD).

#### 3 INVESTIGATIONAL PLAN

# 3.1 Overall Study Design and Plan

This is a multicenter randomized, double-blind, placebo-controlled parallel assignment study followed by an open-label extension (OLE) period. Patients will be randomized to two groups (2:1, Group A or B) and will receive subcutaneous (SC) SA237 (Group A) or placebo (Group B) at Weeks 0, 2, 4, and every 4 weeks (Q4W) thereafter. The randomization will be stratified by prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others) and the most recent attack in the last one year prior to screening (first attack or relapse). If a patient was administered B-cell depleting therapies (e.g. anti-CD20 antibody [e.g. rituximab], anti-CD19 antibody) at least once in the year prior to baseline, the patient will be stratified into "B-cell depleting therapy group" and otherwise into the "immunosuppressants/others group" (e.g. oral corticosteroids, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, tacrolimus).

Patients who experience a protocol-defined relapse which is adjudicated by the Clinical Endpoint Committee (CEC) in the double-blind period or complete the double-blind period can enter the open-label extension period. The double-blind period of the study ends when the total number of CEC-confirmed protocol-defined relapses is 44. At the end of the double-blind period, the clinical cut-off date for the primary analysis will be on the day of the onset of the protocol defined 44<sup>th</sup> relapse (adjudicated by the CEC) or 1.5 years after the date of randomization of the last patient enrolled, whichever comes first. In the extension period, patients can receive open-label treatment with 120 mg SA237 SC at Weeks 0, 2, 4, and every 4 weeks (Q4W) thereafter, until commercial availability of SA237 or Sponsor's decision to discontinue the development program.

For patients who experience a relapse in the double-blind period, appropriate rescue therapy for relapse will be administered. For patients who experienced a relapse which is adjudicated by the CEC as a protocol-defined relapse, SA237 should start under stable disease conditions (i.e. Day 31 or later, where Day 1 is defined as the day of onset of a protocol-defined relapse confirmed by CEC). For patients who completed the double-blind


Related to: SOP-GDO-WW-019 

period of the study. SA237 should start after 4 weeks from the last dosing in the doubleblind period.

The extension period is expected to last until the Last Observation Visit.

Those patients who experience 2 relapses in the extension period, both with a more severe intensity than the last relapse prior to baseline must be discontinued from treatment. It is the investigator's decision whether the patient can continue in the extension period. If the relapses are not as severe as the relapse prior to baseline they can remain in the extension period without being limited to the total number of relapses.

Figure 1 **Study Design** 



Patients who withdraw from the study treatment in the double-blind period due to a clinical relapse should be asked to continue into the Safety Follow Up (SFU) period, which will last for 24 weeks from the last dose of SA237 or placebo.

#### 3.2 Efficacy and Safety Variables

# 3.2.1 Efficacy Variables

The primary efficacy variable is the time to first protocol-defined relapse (TFR) based on CEC evaluations. TFR is defined as the time from the date of the randomization until the first occurrence of relapse (day of onset as reported by the investigator) throughout the double-blind period.

The secondary efficacy variables include change in Visual Analogue Scale (VAS) for pain score, change in Functional Assessment Of Chronic Illness Therapy (FACIT) Fatigue scale score, change in Short Form generic health survey (SF-36) score, change in EQ-5D score, change in Timed 25-Foot Walk (T25W) score, proportion of relapse-free patients, annualized relapse rate (ARR), change in modified Rankin Scale (mRS) score, change in Zarit Burden Interview (ZBI) score, change in Expanded Disability Status Scale (EDSS)

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019


score, change in visual acuity (Snellen chart) score, and change in low-contrast visual acuity (Low-contrast Sloan letter chart [LCSLC]) score.

# 3.2.2 Safety Variables

The safety variables include incidence and severity of adverse events (AEs), adverse events of special interest (AESIs), SAEs, injection related reactions (IRRs), injection site reactions (ISRs), patient withdrawals due to AEs, vital signs (temperature, systolic blood pressure [SBP] and diastolic blood pressure [DBP] and pulse rate), physical examinations, clinical laboratory tests (hematology, chemistry, and urinalysis), 12-lead ECG, body weight, and suicidality (Columbia-Suicide Severity Rating Scale [C-SSRS]).

#### 4 STATISTICAL METHODS

## 4.1 Data Quality Assurance

All tables, figures and data listings to be included in the report will be independently checked for consistency, integrity and in accordance with standard PAREXEL procedures.

#### 4.2 General Presentation Considerations

The analyses periods are defined as follows:

- Study duration of double blind period for efficacy analysis
  - Study duration of double-blind period starts on the day of the randomization. The double-blind period ends on the earliest day of 1) clinical cutoff date (CCOD), 2) the day before the first treatment in the extension period, 3) the end of the study, or 4) last contact for patients lost to follow up.
- Double blind period for safety analysis
  - Double blind period starts on the day of first dose of study drug. The double-blind period ends on the same day as the efficacy analysis.
- Study duration of SA237 exposure for safety analysis (for All SA237 analysis)
  - Study duration of SA237 exposure starts on the day of first dose of SA237. Study duration of SA237 exposure ends on the earliest day of 1) CCOD, 2) the end of the study, or 3) last contact for patients lost to follow up.

The definition of summaries by visit is as follows:

- Summaries by visit for double blind period
  - Baseline is defined as the latest data before or on the date prior to first administration with either placebo or SA237. Summarized visits except for baseline are defined as follows. Irregular visits such as unscheduled visit between week X, dose outside the visit window (DOW), extra visit at relapsing, and the end of the study are out of scope. Week X visits are


Related to: SOP-GDO-WW-019

Related to: SOP-GDO-WW-019

directly used for categories of time. In other words, time window is not applied. If there are the same visits data, one representative assessment nearest to the scheduled visit day will be summarized.

- Summaries by visit for All SA237 analysis
  - Baseline is defined as the latest data before or on the date prior to first administration of SA237. Summarized visits except for baseline are defined as follows. Irregular visits such as unscheduled visit between week X, dose outside the visit window (DOW), extra visit at relapsing, and the end of the study are out of scope. Time window is applied as if visit schedules continue in the double-blind period. Middle of each specified day of visit will be used for the range of time window of each visit. One representative assessment nearest to the specified day of visit in time window of each visit will be summarized

Continuous data will be summarized in terms of the mean, standard deviation (SD), median, minimum, maximum and number of observations, unless otherwise stated. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean, median and SD will be reported to one more decimal place than the raw data recorded in the database. In general, the maximum number of decimal places reported shall be four for any summary statistics.

For categorical parameters, the number and percentages of subjects in each category will be presented at the relevant time point. The denominator for percentage will be based on the number of subjects appropriate for the purpose of analysis. Unless otherwise noted, percentages will be presented to one decimal place. Percentages will not be presented for zero counts and 100% will be presented as an integer. The denominator for all percentages will be the number of subjects in that treatment group within the population of interest, unless otherwise noted. Missing category will only be displayed when there are missing data.

For pharmacokinetic endpoints, concentrations will be analyzed using all reported decimal places, and displayed to the same number of decimal places as recorded in the database. If any samples are collected outside of the protocol defined time window (Appendix 1 in the protocol), the relevant values will be excluded for the calculation of descriptive statistics. Furthermore, if the samples are collected more than 6 weeks after the last study drug administration, the relevant values will be excluded for the calculation of descriptive statistics considering the half-life of IgG. Descriptive statistics will include number of the subjects, geometric mean, geometric coefficient of variation (CV) and the 95% confidence interval for the geometric mean of the concentrations, as well as arithmetic mean, SD, median, minimum, and maximum of SA237 concentrations will be calculated by visit and per defined time window post-dose according to the Pharmacokinetics Per-Protocol Set (PK-PPS). The CV will be presented with 1 decimal place. For the calculation of descriptive statistics, a serum concentration below limit of quantification will be substituted by half of lower limit of quantification (i.e. LLOQ/2). If more than half of the measured values are BLQ at any blood sampling time point, the statistics will not be tabulated for that time point and will be shown as "N.C.".


For immunogenicity, below rules will be applied to neutralizing antibodies:

- Except baseline measurement, neutralizing antibodies will be assessed only if anti-SA237 antibody results are positive.
- If SA237 concentration is over 1 ug/mL, the data of the neutralizing antibodies will be excluded for the calculation of descriptive statistics. High concentrations of SA237 could lead to false negative results in the neutralizing antibody analysis

Changes from baseline in categorical data will be summarized using shift tables where appropriate.

P-values greater than or equal to 0.001, in general, will be presented to three decimal places. P-values less than 0.001 will be presented as "<0.001".

Confidence intervals will be presented to one more decimal place than the raw data.

The Confidence Interval for hazard ratio will be calculated based on the Wald type and the relapse rate Confidence Interval will be provided using Kaplan Meier method with a LOGLOG transformation.

All report outputs will be produced using SAS® version 9.2 or a later version in a secure and validated environment.

# 4.3 Handling of Missing dates

Medications with a missing start date, whose stop date is either unknown or after the date of the first dose of study drug, will be considered concomitant. Medications with a missing start date, whose stop date is prior to the date of the first dose of study drug, will be considered as prior medications.

Where the adverse events start dates of year part are missing then the value will not be imputed. For the partial missing situation (month or day missing), the value will be imputed for the analysis purpose.

| Missing pattern | Start Date / Pre-Dosing | End Date / Post-Dosing |
|---|---|---|
| completely missing | leave missing | |
| missing year | leave missing | |
| missing month | set to 'JAN' | set to 'DEC' |
| missing day | set to '01' | set to last day of the month |
| missing month and day | set to '01JAN' | set to '31DEC' |
| missing time | set to '00:00:00' | set to '23:59:59' |
| (concomitant | missing hours: 0 | missing hours: 23 |
| medication) | missing minutes: 0 | missing minutes: 59 |
| | missing seconds: 0 | missing seconds: 59 |
| missing time | set to '23:59:59' | |
| (adverse event) | missing hours: 23 | |
| | missing minutes: 59 | |
| | missing seconds: 59 | |

These rules apply to AE and concomitant medication. For AE, beginning/end date of AE, first date of study treatment and date of death are considered to avoid inconsistency.

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019


For Visit data other than efficacy, only missing time rules apply. For efficacy visit data, no imputation is made. For birth date, set missing month to '06' and/or set missing day to '15'.

# 4.4 Study Subjects

# 4.4.1 Disposition of Subjects

Summary tables of subject disposition will be provided as follows:

- A summary table of the number of subjects who were randomized to study treatment, number of subjects receiving at least one dose of study drug, number of subjects ending the double-blind period, number of withdrawals from the double-blind period, reason for withdrawal in the double-blind period, number of subjects entering the safety follow-up after double-blind period, number of subjects finishing the safety follow-up after double-blind period, number of subjects entering the open-label extension period, number of withdrawals from the extension period, reason for withdrawal in the extension period, number of subjects conducting last observation visit or withdrawal visit will be provided by treatment group and overall for both the double-blind and the open label extension period.
- A by-subject listing of disposition status, including the date of informed consent, date
  of treatment with study drug and study completing/withdrawal, and reason for
  withdrawal from treatment.

#### 4.4.2 Protocol Deviations

Major protocol deviations are defined as those deviations from the protocol likely to have an impact on the subject's rights, safety, well-being, and/or on the validity of the data for analysis. The impact of major protocol deviations on the efficacy results will be investigated by assessing the robustness of the study results and conclusions to the choice of analysis population (ITT vs per-protocol population, see Section 4.5),

A summary table and listing of protocol deviations will be provided as follows:

- The number and percentage of subjects without any major deviation, with at least 1
  major protocol deviation, and type of major protocol deviations will be summarized by
  randomized treatment group, overall and by site. (Analysis population: All
  Randomized Subjects)
- A by-subject listing of major protocol deviations will be presented. (Analysis population: All Randomized Subjects)

## 4.5 Analysis Populations

The intent-to-treat (ITT) population consists of all randomized subjects and will serve as the primary population for the analysis of efficacy. Subjects will be analyzed as randomized for analysis purposes. In case a patient is incorrectly stratified at time of randomization the analysis will be performed as stratified during randomization.

The Per-Protocol Set population (PPS) will include all patients in the ITT population who

received at least 3 doses of study drug, and without any major protocol deviations which are considered to have an impact on efficacy. Subjects will be analyzed as treated for analysis purposes in the PPS.

The Safety Set (SAF) population will include all randomized subjects who have received at least one dose of active study drug or placebo. Subject will be included in the treatment group corresponding to the trial treatment they actually received for the analysis of safety data using the SAF population, i.e. patients who received at least one dose of SA237 will be assigned to the SA237 treatment arm, irrespective of randomized arm.

The All-Subjects-Treated (All SA237) population will be defined as all enrolled subjects who took at least one dose of active study drug at any time. Date of the first active study drug administration will be defined as Day 1 for All SA237 analysis (i.e. Day 1 of subjects randomized to the placebo group is redefined on the day of first dose of SA237 when entering extension period.

The Pharmacokinetics Per-Protocol Set (PK-PPS) and immunogenicity (anti-SA237 antibody) will include all subjects in the SAF with at least 1 valid post-dose concentration result with a dosing record and sampling time. Pharmacodynamics variables will be analyzed using the SAF population.

The following summary and listing will be provided based on all randomized subjects:

- A summary of analysis populations, including the number and percentage of subjects in the defined analysis sets by treatment group and overall.
- A by-subject listing of analysis population (ITT, PPS, SAF, All SA237 and PK-PPS) information will be provided.

This listing should include: subject number, inclusion/exclusion flag for each population and reason for exclusion from each population.

## 4.6 Demographic and Baseline Characteristics

Summary tables and listing will be provided as follows for ITT, PPS, PK-PPS and SAF.

Demographics and baseline characteristics will be summarized as collected at screening or baseline visit before administration of first dose of study drug and will include:

- gender,
- race (American Indian/Alaska Native, Asian [Japanese], Asian [Non-Japanese], Black/African American, Native Hawaiian/other Pacific Islander, White and Other),
- geographic region (Asia, Europe/other),
- age (years), Age category(<65, >=65 years)
- ethnicity,
- height,
- body weight (the first and the third quartiles of body weight will be presented),
- body mass index (BMI, kg/m2), BMI category ( $<18.5, \ge 18.5$  to  $<25, \ge 25$  to <30, and  $\ge 30$  kg/m2),

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019 

- Prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others),
- Most recent attack in the last one year prior (first attack or relapse),
- AQP4 status at screening (positive, negative), and
- Diagnosis (NMO, NMOSD) by treatment group and overall.

The following listing will be provided.

• A by-subject listing of demographic data.

Age will be calculated as the number of complete years between a subject's birth date and the date of the first informed consent.

# 4.7 Medical History

Medical history will be classified according to the terminology of the latest version of the Medical Dictionary for Regulatory Activities (MedDRA).

Medical conditions are categorized as past or baseline as follows:

- Past diseases: Medical conditions which are specified as start date is before Day 1 Visit date with no ongoing status or the stop date is prior to Day 1 Visit date.
- Baseline diseases: Medical conditions which are specified as start date is before Day 1 Visit date with ongoing status or with the stop date on or after Day 1 Visit date.

The following summaries will be provided by treatment group and overall, based on the SAF.

- A summary table of past diseases will be provided by system organ class (SOC) and preferred term (PT), by treatment group and overall.
- A summary table of baseline diseases will be presented by SOC and PT, by treatment group and overall.
- A by-subject listing of medical history data will be provided.

#### 4.8 Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD).

Medication start and stop dates will be compared to the date of the first dose of randomized study drug and thus the medications will be classified as Prior and / or Concomitant.

Medications that start and stop prior to the date of first dose of study drug will be classified as Prior medications. Medications taken on or after (including ongoing) the first dose of study drug will be classified as Concomitant medication. If a medication starts before the date of first dose of study medication and stops on or after the date of first dose of study medication then the medication will be classified as both Prior and Concomitant medication. NMO/NMOSD pain drugs will be reported as collected on the CRF.


Related to: SOP-GDO-WW-019 

- A summary table of Prior Medications (other treatments than NMO/NMOSD) will be provided by anatomical therapeutic chemical (ATC) and PT.
- A summary table of Concomitant Medications (other treatments than NMO/NMOSD) will be provided by ATC and PT.
- A summary table of Prior NMO/NMOSD drugs for relapse prevention will be provided by ATC and PT.
- A summary table of Concomitant NMO/NMOSD drugs for relapse prevention will be provided by ATC and PT.
- A summary table of Prior NMO/NMOSD drugs for relapse/rescue therapy will be provided by ATC and PT.
- A summary table of Concomitant NMO/NMOSD drugs for relapse/rescue therapy will be provided by ATC and PT.
- A summary table of Prior NMO/NMOSD pain drugs will be provided by ATC and PT.
- A summary table of Concomitant NMO/NMOSD pain drugs will be provided by ATC and PT.
- A summary table of Prior other NMO/NMOSD drugs will be provided by ATC and PT.
- A summary table of Concomitant other NMO/NMOSD drugs will be provided by ATC and PT.
- A by-subject listing of Prior medication data will be provided for NMO/NMOSD
- A by-subject listing of Concomitant medication for NMO/NMOSD.

### 4.9 Treatment Compliance

Overall compliance will be assessed for each subject. Compliance will be computed by determining the number of SC injections relative to the number of SC injections that should have been administered. The compliance will only be evaluated during the double-blind period. For subjects who experience a protocol-defined relapse which is confirmed by CEC or discontinued from study treatment early, the number of planned and actual SC injections will be counted based on the visits before the discontinuation. Treatment compliance will be summarized in terms of compliance based on the Safety population.

Compliance will be calculated using the following formula:

Compliance (%) = 
$$\frac{\text{Number of SC injections during the double-blind period}}{\text{Number of planned SC injections during the double-blind period}} \times 100$$

The following summaries and listings will be provided:

• A summary table of compliance will be presented by treatment group, and overall. The number and percentage of treatment compliance will also be presented by categorized compliance as: <80%, 80%-100%, >100%.


Related to: SOP-GDO-WW-019


 A by-subject listing of study drug administration as well as overall compliance during study duration of the double blind and study duration of the SA237 exposure

# 4.10 Efficacy Evaluation

For the definition of the double-blind period for efficacy evaluations see section 4.2. See Appendix 7.1 how to describe models with SAS code.

### 4.10.1 Analysis and Data Conventions

This study is designed to assess the efficacy of SA237 over placebo in the treatment of NMO/NMOSD. The null hypothesis for primary endpoint will be that there is no difference on the TFR between SA237 monotherapy and placebo during the double-blind period. The alternative hypothesis will be that there is a difference in TFR during double-blinded period.

A two-sided stratified log-rank test at 5% level will be used to test this hypothesis.

#### 4.10.1.1 Multi-center Studies

For the purpose of the summaries and analyses, the term 'Center' will be used to define each site.

All centers will be pooled for the purpose of analysis.

Descriptive summaries will not be presented by individual center. Patient data listing will be provided by individual center.

## 4.10.1.2 Adjustments for Covariates

The primary efficacy analysis will be adjusted for the following baseline covariates:

- Prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others)
- Most recent attack in the last one year prior to screening (first attack or relapse).

For each covariate, a statistical test for the presence of a treatment-by-covariate (i.e. stratification factors) interaction will be performed, by including the interaction term in the secondary analysis model. Subgroup analyses will be performed to further explore the treatment-by-covariate interactions. If any of the treatment-by-covariate are found to be statistically significant, conclusions based on the secondary analysis (no interaction) will be interpreted with caution.

In addition, the ANCOVA and the Mixed-effect model repeated measures (MMRM) for secondary endpoints will be adjusted for prior therapy for prevention of NMO/NMOSD attack and most recent attack in the last one year prior to baseline (stratification factors).

## 4.10.1.3 Handling of Dropouts or Missing Data


For details on censoring rule for the primary endpoint, see section 4.10.2 and handling of missing data for the key secondary efficacy endpoints see section 4.10.3.

For secondary continuous endpoints, a Mixed-effects model repeated measures analysis incorporating all data in double blind period will be used to utilize all the data collected over time with consideration of the variance-covariance matrix of the repeated measures. This method allows a general unstructured variance-covariance matrix and will include data from patients with incomplete data from some scheduled time points.

For FACIT fatigue questionnaire, if there are less than 7 responses recorded, then the total fatigue score will be considered missing. If there are 7 or more responses recorded, then the total fatigue score for that questionnaire will be calculated as the average of the non-missing scores multiplied by 13.

## 4.10.1.4 Multiple Comparisons/Multiplicity

The serial gatekeeping methodology will be employed to control the rate of false positive for the primary endpoint (TFR based on CEC confirmed protocol-defined relapses) and key secondary endpoints (change in VAS for pain to Week 24 and change in the FACIT fatigue scale to Week 24). The 3 efficacy endpoints will be analyzed in hierarchical order, beginning with the TFR based on protocol-defined relapses, followed by the VAS for pain, and ending with FACIT fatigue. A fixed-sequence approach will be applied to control the overall significance level at 0.05. An initial null hypothesis will be tested for the first hierarchical primary efficacy endpoint, the TFR based on protocol-defined relapses. If this is significant, then a repeat of the aforementioned testing procedure for the second hierarchical key secondary endpoint, the VAS for pain will be done. This will be repeated a third time for the FACIT fatigue if the VAS for pain showed a significant difference.

## 4.10.1.5 Examination of Subgroups

The primary and key secondary endpoints (TFR, change from baseline to week 24 in pain and fatigue) will be summarized by the following subgroups:

- NMO/NMOSD and AQP4 Status at screening (5 categories: NMO, NMOSD, NMO and AQP4 positive, NMO and AQP4 negative, and NMO/NMOSD and AQP4 positive)
- Geographical region (Asia, Others).
- Prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others)
- Most recent attack in the last one year prior to screening (first attack or relapse).
- ADA status (ADA negative subjects, ADA unaffected subjects, Treatment-boosted ADA subjects, Treatment-induced ADA subjects) (see Section 4.13)

#### 4.10.1.6 EQ-5D Scoring Algorithm

The EQ-5D 3 level version (EQ-5D 3L) descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problem, some problems, and extreme problems. The


Related to: SOP-GDO-WW-019 

scoring algorithm (US) as described in appendix 7.2 will be used but other norms may be explored for sensitivity analysis.

The EQ-5D index score will be missing in case any answer to one of the five EQ-5D dimensions is missing.

The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale ranging from 0 to 100 where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.

## 4.10.1.7 SF-36 Scoring Algorithm

The SF-36 is a multi-purpose, short form health survey with 36 questions. It yields an 8-scale profile (vitality, physical functioning, bodily pain, general health, role-physical, role-emotional, social role functioning and mental health) of functional health and well-being scores as well as psychometrically based physical and mental health summary measures and a preference based health utility index.

The SF36 will be scored using the Quality Metric proprietary scoring system (version 4.5). Component and domain scores are transformed to a 0-100 scale based on the 2009 US Normative population. Higher scores are indicative of better health related quality of life and a score of 50 is average for the US population.

For the SF-36, missing data rules will be applied according to the proprietary scoring software provided by the license holder (Maruish et al. 2011 p57 and p60).

# 4.10.1.8 FACIT-Fatigue Scale Scoring Algorithm

The FACIT Fatigue scale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. As each of the 13 items of the scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best. Items are scored as follows: 0 = Not at all; 1= A little bit; 2= Somewhat; 3= Quite a bit; 4= Very much. All items are reverse scored except item An5 (*I have energy*) and An7 (*I am able to do my usual activities*). See Table 5-1 for further guidance.

When there are missing data, a total score is prorated from the score of the answered items, as long as more than 50% of the items are answered (i.e. a minimum of 7 of 13 items). The prorated score is calculated as the average of the non-missing scores multiplied by 13.

Table 5-1: FACIT scoring

| Item code | Reverse iter | n Item response | Item score |
|-----------|--------------|-----------------|-------------|
| HI7 | 4 - | | |
| HI12 | 4 - | = | |
| An1 | 4 - | | |
| An2 | 4 - | = | |
| An3 | 4 - | = | <del></del> |
| An4 | 4 - | = | |
| An5 | 0 + | | |
| An7 | 0 + | = | |

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019 Confidential Version 7.0 Version Date: 28NOV2018


| An8 | 4 | - | = | _ |
|---|---|---|---|---|
| An12 | 4 | _ | = | |
| An14 | 4 | _ | = | |
| An15 | 4 | _ | = | |
| An16 | 4 | - | | |
| | | Multiply by | dual item scores: v13: number of items answered: | =FACIT |

#### 4.10.1.9 **EDSS Scoring**

The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurological exam) to 10 (death due to NMO) in 0.5 unit increments that represent higher levels of disability. The EDSS scoring will be based on the score recorded on CRF.

#### 4.10.1.10 mRS Scoring

The mRS is a 7-point disability scale that assesses the degree of disability in patients with neurological impairment. Possible scores range from 0 (no symptom at all) up to 6 (death). The higher scores reflect increased disability. The mRS scoring will be based on the score recorded on CRF

#### 4.10.1.11 **ZBI Scoring**

The ZBI is the measurement to assess caregiver burden. The 22 items ask for the strain caregivers perceive. Responses range from 0 (never) to 4 (nearly always) with maximum score of 88. The higher the total score, the heavier the perceived burden. The ZBI scoring will be based on the score recorded on CRF. For summary tables, only questionnaire with responses to 17 or more out of 22 questions ( $\geq$ = 75% valid response) are used.

The ZBI can be scored if 17 or more items are completed. Interpretation approach can be used if at least 75% of the items have been completed:

- Sum the items that were answered.
- Divide the sum by the number of items that were answered to yield the mean response per item.
- Multiply the mean response per item by 22 (the total items in the scale).

#### 4 10 1 12 Visual acuity function (Snellen chart)

Visual acuity will be measured by a Snellen 20-foot wall chart. The test will be performed monocularly and subjects may use their habitual distance glasses or contact lenses. If visual acuity is less than 20/200, these data will be recorded on CRF as below:

- If the subject can count fingers, this is recorded as "20/300" (CF).
- If the subject can see finger movements, this is recorded as "20/400" (HM).
- If the subject can perceive the flashlight, this is recorded as "20/500" (LP).
- If the subject cannot perceive the flashlight, this is recorded as "20/600" (NLP).

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019


In order to calculate change from baseline, visual acuity scores will be converted to logMAR visual acuity scoring. Transformation of scores will be conducted based on the following table (Table 5-2). If the record of visual acuity score (Snellen chart) is worse than 20/200 (i.e. CF, HM, LP or NLP in this study), the score will be converted to logMAR 1.85, logMAR 2.00, logMAR 2.70 and logMAR 3.00, respectively. If a score which is not in the table is recorded, it would be adjusted to the following lower score (e.g. 20/27 will be converted to 20/30).

Table 5-2: logMAR visual acuity scoring

| Snellen chart | LogMAR |
|---------------|--------|
| 20/10 | -0.30 |
| 20/12.5 | -0.20 |
| 20/15 | -0.12 |
| 20/16 | -0.10 |
| 20/20 | 0.00 |
| 20/25 | 0.10 |
| 20/30 | 0.18 |
| 20/32 | 0.20 |
| 20/40 | 0.30 |
| 20/50 | 0.40 |
| 20/60 | 0.48 |
| 20/63 | 0.50 |
| 20/70 | 0.54 |
| 20/80 | 0.60 |
| 20/100 | 0.70 |
| 20/114 | 0.76 |
| 20/125 | 0.80 |
| 20/150 | 0.88 |
| 20/160 | 0.90 |
| 20/200 | 1.00 |
| CF | 1.85 |
| HM | 2.00 |
| LP | 2.70 |
| NLP | 3.00 |

## 4.10.2 Primary Efficacy Variable

The primary efficacy analyses will be based on the ITT population. Supportive evaluations will be performed using the PPS population.

The primary efficacy endpoint is TFR based on protocol-defined relapses confirmed by the CEC with EDSS/FSS assessment performed by the examining assessor within 7 days after relapse symptoms were reported to the site by the subject. TFR is defined as the time from the date of the randomization until the first occurrence of relapse throughout the double-blind period. Time point of relapse onset is defined as time at which the subject

TP-GDO-WW-016-01 Confidential Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019

Version 7.0

experiences any new or worsening neurological NMO/NMOSD symptoms representing clinical relapse(s) which is later confirmed by the CEC as protocol-defined.

Patients will be censored at the end of double blind period for efficacy analysis (see section 4.2).

The primary analysis of the study is to test the equality of the TFR distribution between the SA237 and Placebo arms:

$$H_0$$
: TFR<sub>SA237</sub> = TFR<sub>placebo</sub> versus  $H_1$ : TFR<sub>SA237</sub>  $\neq$  TFR<sub>placebo</sub>

A stratified log-rank test using strata of prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others) and the most recent attack in the last year prior to baseline (first attack or relapse) will be used.

The Kaplan-Meier method will be used to estimate the TFR based on protocol-defined relapse distribution for each treatment group. The Kaplan-Meier curve will provide a visual description of the differences across treatment groups. In addition, estimates of the treatment effect will be expressed as hazard ratio and 95% confidence intervals using a Cox proportional-hazards model (Exact method will be used for tie data). The model will be stratified by prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others) and the most recent attack in the last one year prior to screening (first attack or relapse). Treatment by covariate interactions will be assessed by including the pairwise interaction terms in the Cox proportional-hazards model.

The following summary tables, figures and analyses will be provided for the ITT and PPS:

- A summary table of Kaplan-Meier estimate of TFR (protocol-defined relapse) will be presented by treatment group.
- A figure of Kaplan-Meier estimate of TFR (protocol-defined relapse) will be presented by treatment group.
- Analysis of TFR (protocol-defined relapse) will be performed using stratified log-rank test.
- Analysis of TFR (protocol-defined relapse) will be performed using stratified Cox regression.

TFR (protocol-defined relapse) will be presented for the subgroups defined in section 4.10.1.5.

Additionally, sensitivity analyses of TFR (protocol-defined relapse) using a weighted stratified log-rank test, TFR (clinical relapse), TFR (treated clinical relapse), TFR (treated clinical relapse: optic neuritis), and protocol-defined relapse based on CEC adjudication (regardless of assessment limit of 7 days) will be conducted for ITT as follows For all sensitivity analyses, the same strata as for the primary endpoint will be used.

TFR (protocol-defined relapse) using a weighted stratified log-rank test: The sample size assumptions include a delayed treatment effect (see section 4.14). The influence of a

Effective Date: 28Aug13 Version Date: 28NOV2018
Related to: SOP-GDO-WW-019 

potential delayed treatment effect will be assessed by using a weighted log-rank test using Fleming-Harrington weight function. Treatment effect is estimated adjusting for a change in the hazard ratio over time (i.e. non-proportional hazards). Based on simulations using blinded SA309 data, the parameters of the weight function are set to be rho=0 and gamma=1 (Lee 2007).

Clinical relapses: All relapses reported by investigators will be handled as events for TFR

Treated clinical relapses: Relapses treated with rescue therapy will be handled as events

Treated clinical relapse: optic neuritis: Relapses treated with rescue therapy and judged as optic neuritis by the investigator will be handled as events.

Optic neuritis will be identified via relapse assessment form before data base lock (for details see appendix 7.3). The same censoring rules as for the primary endpoint will be applied, except for the specific event of interest.

TFR (protocol-defined relapse) censored by affecting medications: Censored at the first timing of the start date of following medications:

- 1. Relapse prevention therapy
- 2. Rescue therapy
- 3. Systemic administration of steroid for other indication for more than 5 days
- A summary table of Kaplan-Meier estimate of TFR (clinical relapse) will be presented by treatment arm.
- A summary table of Kaplan-Meier estimate of TFR (treated clinical relapse) will be presented by treatment arm.
- A summary table of Kaplan-Meier estimate of TFR (treated clinical relapse: optic neuritis) will be presented by treatment arm.
- A summary table of Kaplan-Meier estimate of TFR (protocol-defined relapse based on CEC adjudication, regardless of assessment limit of 7 days) will be presented by treatment arm.
- A summary table of Kaplan-Meier estimate of TFR (protocol-defined relapse) censored by affecting medications will be presented by treatment group.
- A figure of Kaplan-Meier estimate of TFR (clinical relapse) will be presented by treatment group.
- A figure of Kaplan-Meier estimate of TFR (treated clinical relapse) will be presented by treatment group.
- A figure of Kaplan-Meier estimate of TFR (treated clinical relapse: optic neuritis) will be presented by treatment group.

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019

- A figure of Kaplan-Meier estimate of TFR (protocol-defined relapse based on CEC adjudication, regardless of assessment limit of 7 days) will be presented by treatment group.
- A figure of Kaplan-Meier estimate of TFR (protocol-defined relapse) censored by affecting medications will be presented by treatment group.
- Analysis of TFR (protocol-defined relapse) will be performed using a weighted stratified log-rank test and the parameters of the weight function are set to be rho=0 and gamma=1.
- Analysis of TFR (clinical relapse) will be performed using stratified log-rank test.
- Analysis of TFR (treated clinical relapse) will be performed using stratified log-rank test.
- Analysis of TFR (treated clinical relapse: optic neuritis) will be performed using stratified log-rank test.
- Analysis of TFR (protocol-defined relapse based on CEC adjudication (regardless of assessment limit of 7 days)) will be performed using stratified log-rank test.
- Analysis of TFR (protocol-defined relapse) censored by affecting medications will be performed using stratified log-rank test.
- Analysis of TFR (clinical relapse) will be performed using the stratified Cox regression.
- Analysis of TFR (treated clinical relapse) will be performed using the stratified Cox regression.
- Analysis of TFR (treated clinical relapse: optic neuritis) will be performed using the stratified Cox regression.
- Analysis of TFR (protocol-defined relapse based on CEC adjudication (regardless of assessment limit of 7 days)) will be performed using the stratified Cox regression.
- Analysis of TFR (protocol-defined relapse) censored by affecting medications will be performed using stratified Cox regression.
- A by-subject listing of TFR, which also includes clinical relapse, treated clinical relapses and treated clinical relapse: optic neuritis, will be provided.

# 4.10.3 Secondary Efficacy Variables

The key secondary efficacy endpoints are change from baseline in VAS for pain score and the FACIT fatigue scale score to week 24. All efficacy analyses will be based on the ITT population and the double-blind period.

### 4.10.3.1 Key Secondary Endpoints

 Analysis of change in VAS for pain score from baseline to week 24 using ANCOVA (BOCF).


Related to: SOP-GDO-WW-019 

• Analysis of change in FACIT fatigue scale score from baseline to week 24 using ANCOVA (BOCF).

The ANCOVA will include treatment group as fixed effect; the baseline measurements and stratification variables as covariates.

The missing data will be imputed by baseline observation carried forward (BOCF) method.

Additionally, sensitivity analyses using different imputation methods (random hot deck, imputation using OLE baseline/withdrawal visits) and MMRM using all collected data during the double-blind period will be performed as follows:

#### Random hot deck:

Random hot deck imputation method using a regression based approach will be conducted. In this imputation method, missing values will be replaced with values from a similar responding unit.

Imputation using OLE baseline/ withdrawal visits:

VAS for Pain and fatigue are assessed at OLE baseline visit for patients entering into OLE and the withdrawal visit for patients discontinuing from treatment. Missing values for patients that do not have a Week 24 assessment, but for which a pain /fatigue assessments is available between study days 85 and 252 from an OLE baseline or withdrawal visit, will be replaced with these values. The remaining missing values will be imputed using BOCF.

- Analysis of change in VAS for pain score from baseline to week 24 using ANCOVA by random hot deck imputation method.
- Analysis of change in FACIT fatigue scale score from baseline to week 24 using ANCOVA by random hot deck imputation method.
- Analysis of change in VAS for pain score from baseline to week 24 using ANCOVA with imputation using OLE baseline/ withdrawal visits
- Analysis of change in FACIT fatigue scale score from baseline to week 24 using ANCOVA with imputation using OLE baseline/ withdrawal visits

The following summary tables and analyses including all available visits in the double-blind period will also be provided as exploratory analyses:

- A summary table of change in VAS for pain score from baseline to every 24 weeks.
- A summary table of change in FACIT fatigue scale score from baseline to every 24 weeks.
- Analysis of change in VAS for pain score from baseline to every 24 weeks using MMRM analysis.


Analysis of change in FACIT fatigue scale score from baseline to every 24 weeks using MMRM analysis.

The MMRM will include treatment group, protocol-specified visit, treatment-by-visit interaction as fixed effects; the baseline measurements and stratification variables as covariates: and visit as a repeated measure. The unstructured covariance matrix will be assumed in the model

If the unstructured covariance matrix does not converge, the length of the observation interval will be limited (e.g. to Week 96) and/or other covariance structure will be used. If treatment-by-visit interaction is not statistically significant, the full model will be kept.

If the normality assumption for the key secondary variable does not hold, GEE or Generalized Linear Mixed-effect model analysis will be used. The assessment will be performed prior to unblinding.

#### 4.10.3.2 Other Secondary Endpoints

The following summary tables, figures and analysis will be provided for the ITT:

- A summary table of change in SF-36 domain scores from baseline to every 24 weeks.
- A summary table of change in SF-36 summary score (physical and mental) from baseline to every 24 weeks.
- A summary table of change in EQ-5D scores from baseline to every 24 weeks.
- A summary table of change in T25W from baseline to every 24 weeks.
- A summary table of the proportion of relapse-free patients.
- A summary table of ARR.

The ARR is calculated as the total number of relapses experienced divided by the person-years at risk. The 95% CI will be presented based on the Poisson distribution. ARR based on the person-years at risk on the total study period will also be provided. In order to account for different study treatment exposure durations among subjects, log-transformed exposure time will be included in the model as an "offset" variable for appropriate computation of ARR.

- A summary table of ARR for patients with clinical relapse.
- A summary table of ARR for patients with treated clinical relapse.
- Analysis of ARR will be performed using negative binomial regression model (protocol-defined relapse).

For comparing the difference between 2 treatment arms, relapse number will be the response variable; treatment group, prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others) and the most recent attack in the last one year prior to baseline (first attack or relapse) as covariates. Logtransformed exposure time will be included in the model as an "offset" variable.

A summary table of change in mRS scores from baseline to every 24 weeks.

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019

- A summary table of change in ZBI scores from baseline to every 24 weeks.
- A summary table of change in EDSS scores from baseline to every 24 weeks.
- A summary table of change in visual acuity (Snellen chart) scores from baseline to every 24 weeks.
- A summary table of change in low-contrast visual acuity (Low-contrast Sloan letter chart [LCSLC]) scores from baseline to every 24 weeks.
- Analysis of change in SF-36 domain scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in SF-36 components (physical and mental) from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in EQ-5D scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in T25W scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in mRS scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in ZBI scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in EDSS scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in visual function (Snellen chart) scores from baseline to every 24 weeks using MMRM analysis.
- Analysis of change in low-contrast visual acuity (Low-contrast Sloan letter chart [LCSLC]) scores from baseline to every 24 weeks using MMRM analysis.

The MMRM will include treatment group, protocol-specified visit, treatment-by-visit interaction as fixed effects; the baseline measurements and stratification factors as a covariate; and visit as a repeated measure. The unstructured covariance matrix will be assumed in the model.

If the unstructured covariance matrix does not converge, the length of the observation interval will be limited (e.g. to Week 96) and/or compound symmetric structure will be used. If treatment-by-visit interaction is not statistically significant, the full model will be kept.

If the normality assumption for other secondary variables does not hold, GEE or Generalized Linear Mixed-effect model analysis will be used. The assessment will be performed prior to unblinding.

### **4.11 Safety Evaluation**


Related to: SOP-GDO-WW-019


Unless otherwise specified, all safety summaries and analyses will be based upon the SAF as defined in Section 4.5

## 4.11.1 Subgroup analyses

Main safety data will be summarized by the same subgroups as for the efficacy analyses (see section 4.10.1.5). Baseline weight (<median, >= median) will be included in addition.

# 4.11.2 Extent of Exposure

Duration of exposure to study drug (days) is defined as date of last dose - date of first dose + 1, and will be summarized.

The following exposure summaries will be produced:

- A summary of exposure duration and study duration (days).
- A summary of the number of doses and total cumulative dose of study drug.

#### 4.11.3 Adverse Events

Adverse events will be coded using MedDRA. All summaries will be sorted alphabetically by System Organ Class (SOC) and preferred term (PT), starting with the most frequent event. All adverse events reported in whole study will be reported in listings. For AEs, if the AE intensity is missing, the worst case (severe) will be assumed. If the drug relationship is missing, the worst case (drug related) will be assumed. In summaries, multiple occurrences of the same PT event in one individual will be counted only once.

The following summary tables of AEs will be provided:

- An overall summary of AEs will be presented. It will include the number and percentage
  of subjects with at least 1 AE, serious AE, AE leading to early discontinuation, adverse
  drug reaction, and severe AE and number of death.
- A summary of AEs by SOC and PT.
- A summary of AEs by Intensity, SOC and PT.
- A summary of AEs leading to discontinuations of treatment.
- A summary of AEs leading to dose interruption.
- A summary of adverse drug reactions (ADRs) by SOC and PT.
- A by-subject listing of all AEs.
- A by-subject listing of all AEs leading to discontinuation.
- A by-subject listing of all AEs leading to drug interruption.
- A by-subject listing of all ADRs.

TP-GDO-WW-016-01
Effective Date: 28Aug13
Related to: SOP-GDO-WW-019

Confidential Version 7.0 Version Date: 28NOV2018

# 4.11.4 Deaths, Serious Adverse Events, and Other Significant Adverse Events

SAE will be provided by treatment group. SAE will be provided by subgroups The following summary tables of SAEs will be provided:

- A summary of incidence of serious AEs (SAEs) by SOC and PT.
- A summary of incidence of SAEs leading to discontinuation by SOC and PT.
- A by-subject listing for all deaths.

#### 4.11.5 C-SSRS

The following will be presented for C-SSRS:

- A summary of C-SSRS.
- A by-subject listing of C-SSRS.

Scores reported in the "Baseline" and "Prior to study" pages of the CRF will be handled as baseline score. Scores reported in "Since Last Visit" and "Since Study Start" page of CRF will be summarized by visit when the data is recorded.

# 4.11.6 Adverse event of special interest (AESI)

AESI are defined in the protocol as follows and collected in the eCRF using a specific question.

- Cases of an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice.
- Suspected transmission of an infectious agent by the study treatment.

The following listings will be provided:

• A by-subject listing of all AESI.

#### 4.11.5 Selected Adverse Events

## Selected adverse events are

- non serious infections that require treatments with IV antibiotic, antifungal, antiviral
- opportunistic infections defined as per basket with PO antibiotic, antifungal, antiviral injection-related reaction (IRR; an AE which occurs within 24 hours after study treatment injection except where the event is not considered an allergic reaction.

The following summary tables and listings will be provided:

• A by-subject listing for non-serious infection (SOC: Infections and infestations) medicated by IV treatment antibiotic, antifungal, antiviral.

Effective Date: 28Aug13 Version Date: 28NOV2018
Related to: SOP-GDO-WW-019 

 A by-subject listing for opportunistic infection (defined by MedDRA basket in Appendix 7.4) medicated by PO treatment antibiotic, antifungal, antiviral.

# 4.11.7 Infections, Serious Infection,

Serious adverse event in "SOC: Infections and infestations" will be summarized.

Opportunistic infections are defined from all adverse events by MedDRA basket in Appendix 7.4 and reported as described in section 4.11.5 selected adverse events... Serious infection will be provided per 100 patient-years by treatment group during the double-blind period. The patient-years will be based on the double-blind period for safety analysis (see section 4.2). The rate per 100 patient-years by treatment group (along with the 95% CI) will be calculated for serious infections.

The number of serious infections per 100 patient-years is calculated as:

Total number of serious infections / Total number of patient-years ×100

The 95% CI for the number of serious infections per 100 patient-years is calculated as follows:

Exact lower 95% confidence limit = chisq (p = 0.025, df = 2 Y) / (2 T)

Exact upper 95% confidence limit = chisq [p = 0.975, df = 2(Y + 1)] / (2T)

where Y is the total number of serious infections, T is total number of patient-years at risk and chisq (p,df) is the quantile of the upper tail probability of the X2 distribution on df degrees of freedom. This approach has the advantage of providing an estimate for the upper 95% confidence limit even when the total number of serious infections is zero.

The following summary tables will be provided.

- A summary of serious infection by SOC and PT.
- Rates of serious infections by 100 patient-years.
- A by-subject listing of Infections.
- A by-subject listing of Opportunistic Infections.

#### 4.11.8 Anaphylaxis

Anaphylaxis is defined by MedDRA SMQ "Anaphylactic reaction - Narrow" and will be listed

A by-subject listing of Anaphylaxis.

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019


#### **4.11.9 IRR and ISR**

IRR in CRF selected AE (IRR) page will be summarized. ISRs flagged as "Injection site reaction" in CRF selected AE (IRR) or general AE page will be summarized. The following summary tables will be provided:

- A summary of IRR
- A summary of ISRs by SOC and PT.
- A by-subject listing of all IRRs.
- A by-subject listing of all ISRs.

## 4.11.10 Clinical Laboratory Evaluation

For continuous laboratory measurements including hematology, clinical chemistry, and urinalysis, summary using descriptive statistics of the actual values and their change from baseline will be presented by treatment group at each visit. The laboratory tests to be performed are presented in Table 4-4.

When analyzing categorical data, the number and percentage of subjects in each category will be presented. In addition, shift tables may be used to evaluate the number and percentage of subjects having a different post-baseline status when compared to their baseline status.

A subject data listing will be provided for all laboratory data. Values outside the normal range will be flagged within the listing. A subject data listing will also be provided for all treatment emergent marked laboratory abnormalities (see Appendix 7.5).

The following summaries, listings and figures will be provided: by treatment group

- A summary of each laboratory parameter in Table 4-4 and change from baseline will be provided by visit.
- A shift table based on the normal range for each laboratory parameter will be presented by double-blind period endpoint value relative to baseline by treatment group.
- A by-subject listing of laboratory parameters.

Table 4-4 Laboratory measurements

| Hematology | Clinical chemistry | Urinalysis | Complement |
|---|---|---|---|
| Hematocrit Hemoglobin International normalized ratio (INR) Platelet count Red blood cell (RBC) count WBC count | Sodium Potassium Chloride Calcium Phosphorous Ferritin Blood urea nitrogen (BUN) Creatinine | Glucose<br>Protein<br>Urinary occult blood<br>Urobilinogen | Complement tests<br>(C3, C4 and<br>CH50) |

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019 Confidential Version 7.0 Version Date: 28NOV2018


| Absolute | Total bilirubin |
|------------------|---------------------|
| differential | Fibrinogen |
| count | Total serum protein |
| (neutrophils, | Albumin |
| eosinophils, | ALT |
| lymphocytes, | AST |
| monocytes, | Alkaline |
| basophils, other | phosphatase |
| cells) | Gamma-glutamyl |
| , | transpeptidase (γ- |
| | GTP) |
| | Lactate |
| | dehydrogenase |
| | (LDH) |
| | Total cholesterol |
| | Low density |
| | lipoprotein |
| | cholesterol (LDL) |
| | High density |
| | lipoprotein |
| | Cholesterol (HDL) |
| | Triglycerides |
| | Creatine kinase |
| | (CK) |
| | Ùric acid |

#### 4.11.11 AST and ALT:

AST and ALT will be categorized into four group (>3-5 xULN, 6-10 xULN, 11-20 xULN and 21- xULN) based on maximum post-baseline levels within baseline and post-baseline respectively for each test by maximum post-baseline levels for total bilirubin and alkaline phosphatase (total bilirubin <= 2xULN, total bilirubin > 2xULN, total bilirubin > 2xULN and alkaline phosphatase <= 5xULN). The denominator is the number of subjects with any valid assessment at baseline and post-baseline respectively. Subjects with AST or ALT results fulfilling criteria for more than one category are counted only once, in the category indicating the highest elevation level within baseline and post-baseline.

Summary of AST and ALT Results.

# 4.11.12 Electrocardiograms

For quantitative ECG measurements (heart rate, PR interval, QRS duration, QT interval, and corrected QT intervals using Bazett and Fridericia correction methods), values during the double-blind period will be presented by treatment group for all visits.

The Bazett corrected QT (QTcB) will be calculated as

QTcB=QT/RR $^{0.5}$ , where RR = 60/HR.

The Fridericia corrected OT (OTcF) will be calculated as

QTcF=QT/RR $^{0.33}$ , where RR = 60/HR.

Effective Date: 28Aug13 Version Date: 28NOV2018
Related to: SOP-GDO-WW-019 

The following summaries and listings will be provided for the SAF and all SA237:

- A summary of 12-lead by treatment group at each specified visit.
- The number and percentage of subjects with a QTc (using Bazett and Fridericia corrected) of ≤450ms, >450 to ≤480ms, >480 to ≤500ms, and >500ms will be summarized by treatment group at each specified visit.
- The number and percentage of subjects with a QTc (using Bazett and Fridericia corrected) of an increase from baseline of >0 to ≤30ms, >30 to ≤60ms, and >60ms will be summarized by treatment group at each specified visit.
- The number and percentage of subjects with PR interval values ≤120ms, >120 to ≤220ms, and >220ms, and the number and percentage of subjects with QRS interval values ≤60ms, >60 to ≤120ms, and >120ms will be presented by treatment group at each specified visit.
- A summary of incidence of treatment-emergent abnormality 12-lead ECG findings after start of study drug by treatment group.
- A by-subject listing of abnormal 12-lead ECG data will be provided.

# 4.11.13 Vital Signs, Physical Findings and Other Observations Related to Safety

Noninvasive pulse rate, temperature, systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured at visits with the subject in a sitting position after at least 10 minutes at rest, according to the tabular schedule of study procedures in the protocol. Summary statistics of the actual measurement and their changes from baseline will be presented by treatment group at each specified visit.

In addition, summary statistics for the actual value and change from baseline will be presented by treatment group for all visits during the double-blind period.

Abnormal vital sign criteria as follows:

- diastolic blood pressure [DBP]: <50, >100 mmHg
- systolic blood pressure [SBP]: <90, >160 mmHg
- pulse rate [PR]: <60, >100 bpm
- Temperature: <36.0, >38.0

The following summaries and listings will be provided:

- A summary of pulse rates temperature, blood pressure and change from baseline by treatment group and visit.
- The number and percentage of subjects with abnormal vital signs during double-blind period by treatment group.
- A by-subject listing of vital signs.

#### 4.12 Pharmacokinetics and Pharmacodynamics


Related to: SOP-GDO-WW-019

Version Date: 28NOV2018


The serum SA237 concentrations will be reported using the PK-PPS. The PD variables (IL-6, sIL-6R, hsCRP, anti-AQP4Ab, Plasmablast) will be reported using the SAF population.

To determine concentrations of SA237, serum samples will be drawn at various time points throughout the study. At Week 0, blood specimens for PK and PD samples will be collected prior to first dose administration of study drug (blank value). At other visits, PK and PD samples will be collected along with hematology samples at any time prior to drug administration according to the Schedule of Study assessments.

To support the Japanese BLA, the following reports will be produced. SA237 concentrations and PD variables in serum will be listed and summarized using descriptive statistics (including geometric mean and CV%, arithmetic mean and SD, median, observed maximums and minimums, and sample size). Arithmetic mean ± SD serum concentration-time profile and combined all subjects' serum concentration-time profiles (spaghetti plot) will be plotted using linear and semi-log scale. In addition, individual serum concentration-time profile will be plotted for each subjects using linear and semi-log scale. Summary tables and figures of SA237 concentration and PD variables will be provided as follows:

Concentration of SA237 and PD variables (absolute values as well as change from baseline) in serum will be summarized using descriptive statistics and arithmetic mean  $\pm$  SD serum concentration-time profile will be plotted by following subgroup using linear scale.

Samples that were excluded from the summary statistics will be marked in the listing.

The rule for summary of titer for anti AQP4 antibody status is defined in appendix 7.6.

Summary tables, figures, and listings of SA237 concentration and PD variables will be provided as follows:

- Summaries of concentrations of SA237 by visit will be presented by age category, Japanese/non-Japanese, relapse/no-relapse, ADA status, and overall.
- Summary of concentration of IL-6, sIL-6R, and hsCRP by visit will be presented by age category, Japanese/non-Japanese, relapse/no-relapse and overall in each of treatment group.
- Summary of titer for anti AQP4 antibody status, Plasmablast (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), and Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%) and CD19+ (cells/uL)) by visit will be presented by NMO/NMOSD and AQP4 Status, relapse/no-relapse and overall in each of treatment group.
  - \*Plasmablast and CD19+ cells will be calculated by following equation
    - O Plasmablasts (cells/uL) = CD45+Abs \* Plasmablasts/CD45+ (%)


- $\circ$  CD19+ (cells/uL) = CD45+Abs \* CD19+/CD45+ (%)
- A by-subject listing of concentration of SA237 in serum.
- A by-subject listing of IL-6, sIL-6R, and hsCRP

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019 Version 7.0 Version Date: 28NOV2018

- A by-subject listing of anti-AQP4 antibody (positive/negative and titer)
- Plasmablast (Plasmablasts/CD19+(%), Plasmablasts/CD45+(%), and Plasmablast (cells/uL)), and CD19+ cells (CD19+/CD45+(%) and CD 19+ (cells/uL))
- A by-subject spaghetti plot of concentration for SA237 in serum by subgroup (age category, Japanese/non-Japanese, relapse/no-relapse, ADA status) using linear scale and overall using linear and semi log scale.
- A by-subject spaghetti plot of the absolute value and the change from baseline for concentration of IL-6, sIL-6R, and hsCRP by treatment group using linear and semi log scale.
- A by-subject spaghetti plot of the absolute value for concentration of IL-6, sIL-6R, and hsCRP by subgroup (age category, Japanese/non-Japanese, relapse/no-relapse, ADA status) in each of treatment group using linear scale
- A by-subject spaghetti plot of the absolute value for concentration of IL-6, sIL-6R, and hsCRP by treatment group in each subgroup (relapse/no-relapse, ADA status) using linear scale
- A by-subject spaghetti plot of the absolute value and the change from baseline for titer of anti-AQP4 antibody, Plasmablast (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), and Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%), and CD19+ (cells/uL)) by treatment group using linear and semi-log scale
- A by-subject spaghetti plot of the absolute value for titer of anti-AQP4 antibody, Plasmablasts (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), and Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%), and CD19+ (cells/uL)) by subgroup (NMO/NMOSD and AQP4 Status, relapse/no-relapse) in each of treatment group using linear scale.
- A by-subject spaghetti plot of the absolute value for titer of anti-AQP4 antibody, Plasmablast (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), and Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%), and CD19+ (cells/uL)) by treatment group in each subgroup (NMO/NMOSD and AQP4 Status, relapse/no-relapse) using linear scale.
- An Arithmetic mean  $\pm$  SD plot of concentration for SA237 in serum by subgroup (age category, Japanese/non-Japanese, relapse/no-relapse, ADA status) using linear scale and overall using linear and semi log scale.
- An Arithmetic mean ± SD plot of the absolute value and the change from baseline for concentration of IL-6, sIL-6R, and hsCRP by treatment group using linear and semilog scale.


- An Arithmetic mean ± SD plot of the absolute value for concentration of IL-6, sIL-6R, and hsCRP by subgroup (age category, Japanese/non-Japanese, relapse/no-relapse, ADA status) in each of treatment group using linear scale.
- An Arithmetic mean ± SD plot of the absolute value for concentration of IL-6, sIL-6R, and hsCRP by treatment group in each subgroup (age category, Japanese/non-Japanese, relapse/no-relapse, ADA status) using linear scale
- An Arithmetic mean ± SD plot of the absolute value for titer of anti-AQP4 antibody, Plasmablast (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%) and CD19+ (cells/uL)) by treatment group using linear and semi-log scale
- An Arithmetic mean ± SD plot of the absolute value for titer of anti-AQP4 antibody, Plasmablasts (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%) and CD19+ (cells/uL)) by subgroup (NMO/NMOSD and AQP4 Status, relapse/no-relapse) in each of treatment group using linear scale
- An Arithmetic mean ± SD plot of the absolute value for titer of anti-AQP4 antibody, Plasmablast (Plasmablasts/CD19+ (%), Plasmablasts/CD45+ (%), Plasmablasts (cells/uL)), and CD19+ cells (CD19+/CD45+ (%) and CD19+ (cells/uL)) by treatment group in each subgroup (NMO/NMOSD and AQP4 Status, relapse/no-relapse) using linear scale.
- A by-subject listing of actual doses, date and time of sampling, visit, relative day, and the accession number.
- Scatter plot of anti-AQP4 antibody titer versus plasmablast (Plasmablasts/CD19+ Plasmablasts/CD45+ (%), Plasmablasts (cells/uL)) will be presented at Weeks 0, 2 and 4, 8, 12, 24, and Q24W. When the data of anti-AQP4 antibody is negative, put "1" as a titer for negative samples and replace to "BLQ".
- Scatter plots of serum SA237 concentration versus body weight at weeks 2, 4, Q4W respectively.

## 4.13 Immunogenicity

ADA subgroup using confirmatory sample status are defined as below.

- ADA negative subjects: subjects without positive ADA during study. If sample at baseline is missing and no sample after the baseline is positive, the subject is defined as" ADA negative subjects".
- ADA unaffected subjects: subjects who have pre-existing ADA (POSITIVE at baseline) that was NOT boosted to a higher level after the post dose. "NOT boosted


- to a higher level" means that ADA titer after the baseline is <fourfold than the ADA titer at baseline.
- Treatment-boosted ADA subjects: subjects who have pre-existing ADA that was boosted to a higher level at least one time point after baseline "Boosted to a higher level" means as follow
  - 1) ADA titer after the baseline is greater fourfold than the ADA titer at baseline
- Treatment-induced ADA subjects: subjects who have positive ADA not at baseline but after the baseline. If sample at baseline is missing and at least one sample after the baseline is positive, the subject is defined as" Treatment-induced ADA subjects"

The immunogenicity will be analyzed using the SAF population.

- The numbers and proportions of subjects with positive ADA at baseline will be presented by treatment group and overall.
- The numbers and proportions of ADA negative subjects, ADA unaffected subjects, treatment-boosted ADA subjects, and treatment-induced ADA subjects will be summarized. The numbers and proportions of transient ADA and persistent ADA will be summarized in the treatment-induced ADA subjects.

Transient ADA: 1) Treatment-induced ADA detected only at one sampling time point (excluding the last sampling time point) during the study or 2) treatment-induced ADA detected at two or more sampling time points during the study, where the period between first and last ADA-positive sampling time points is less than 16 weeks, and the subject's last sampling time point is ADA-negative.

Persistent ADA: 1) Treatment-induced ADA detected at two or more sampling time points during the study, where the period between first and last ADA-positive sampling time points is 16 weeks or longer or 2) where the period between first and last ADA-positive sampling time points is less than 16 weeks, and the subject's last sampling time point is ADA-positive or 3) treatment-induced ADA detected only at the last sampling time point.

- > The numbers and proportions of patients with positive/negative anti-SA237 antibodies and neutralizing antibodies will be presented at Week 0 and Q4W in SA237 group by visit.
  - A by-subject listing of anti-SA237 antibody (confirmatory judgment (positive/negative), titer, ratio of peak titer/baseline titer, and ADA subgroup), neutralizing judgment (positive/negative)), and adverse events in the subject having anti-SA237 antibody at least once at any point in time.

## 4.14 Determination of Sample Size

Approximately 90 patients need to be recruited and randomized in a 2:1 ratio to the two treatment groups (SA237 and placebo). The sample size considerations are based on the following assumptions:

• A two-sided log-rank test.

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019 

- At least 80% power at the 5% significance level
- The hazard ratio of SA237 over placebo for an initial 2 months from randomization is 1.0. The hazard ratio after an initial 2 months from randomization is 0.25.
- TFR in the placebo arm following an exponential distribution, with hazard rate for 1 year h(t) = 1.1295.
- A 2-year dropout rate of 10%.

Based on the assumptions, 44 TFR events are needed for the primary analysis. The 90 patients enrolled over 33 months and followed for an additional 5 months will provide 44 TFR events. The primary analysis will be performed once 44 TFR events have been observed. The Sponsor will conduct a blind review of the data including accumulation of events during the double-blind period and may take appropriate action such as to increase the number of patients or to extend the double-blind period based on this blind review.

It has been assumed that the number of relapses will follow a Gamma-Poisson distribution and that the variance/mean ratio will be a constant value of  $\sqrt{2}$ . This distribution was assumed and the ratio was estimated using data from MS trials (Gold et al. 2012; Kappos et al. 2010) because there are no approved medications for NMO and no raw data from patients with this indication are available.

Because the mean ARR of NMO patients is estimated at 0.82 and eligibility criterion 2 says patients at least 1 relapse in last 12 months prior to screening are selected, we calculate the zero-truncated mean of the Gamma-Poisson distribution with the mean of 0.82 and the mean and variance ratio of  $\sqrt{2}$ , then the baseline ARR is estimated at 1.65. The posttreatment ARR in the placebo group in NMO patients with anti-AQP4 positive and negative is estimated as 1.5 and 1.0, respectively (Cree et al. 2015). Given that the proportion of patients who are negative for anti-AQP4 antibody at screening will be capped at 30% of the total number of patients in this study, post-treatment ARR is estimated as 1.35.

Using the proportion of zero under supposed ARR distribution, we estimate the relapse-free rate at a year in placebo group at 32.3%. The relapse-free rate is assumed to follow the exponential distribution with a constant hazard, and then we set the hazard for 1 year of 1.1295 in placebo group.

According to tocilizumab case report in NMO patients, the pre- and post- baseline relapse counts were reduced from total 4 counts per 6 months to 1 count per 6 months. Then the pre- and post- baseline ratio of 0.25 is used as the estimation of the mean ARR ratio of tocilizumab compared with placebo. Under the assumption of ARR and relapse-free rate distribution above, the mean ARR ratio is coincided with the hazard ratio. The primary rationale for the mechanism of anti-IL-6 blockade in NMO/NMOSD is the expected inhibition of the survival of plasmablast followed by a reduction in anti-AQP4 antibody. Given that the reduction in anti-AQP4 antibody is required for prevention of relapse, and considering the half-life of immunoglobulin G, sufficient effectiveness might not be expected for an initial period of a few months even if IL-6 signaling is inhibited immediately. So we have set the hazard ratio of SA237 over placebo at 1.0 for an initial 2 months from randomization and at 0.25 after an initial 2 months from randomization.

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019

Version 7.0 Version Date: 28NOV2018


TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019 Version Date: 28NOV2018


## Changes in the Conduct of the Study or Planned Analysis

### 5.1 Amendment from Ver 1.0 to 2.0

The primary purpose of this SAP amendment is to revise the context to align with the statistical section in the amended protocol.

For TFR, the condition of handling missing data has been added. For patients with protocoldefined relapse based on CEC evaluation, but not performed EDSS/FSS assessment within seven days after the patient reports the symptoms to the site, the TFR will be censored on the date of relapse onset. The sensitivity analysis of protocol-defined relapse based on CEC adjudication has also been added.

## 5.2 Amendment from Ver 2.0 to 3.0

The primary purpose of this SAP amendment is to follow the FDA comments:

For primary endpoint, analysis method has changed to the log-rank based permutation test from stratified log-rank test. For key secondary endpoints of VAS and FACIT, ANCOVA has been added for change from baseline at 24 weeks. For primary and key secondary endpoints, SAS code has been added.

#### 5.3 Amendment from Ver 3.0 to 4.0

The primary purpose of this SAP amendment is to revise the context to align with the amended protocol version 5.0 dated 5 Nov 2015. For TFR, the definition of censoring has been revised.

#### 5.4 Amendment from Ver 4.0 to 5.0

The primary purpose of this SAP amendment is to revise the context to align with the amended protocol version 6.0 dated 1 March 2016. The assumption for determination of sample size has been revised. For key secondary endpoints, sensitivity analysis has been added

#### 5.5 Amendment from Ver 5.0 to 6.0

The primary purpose of this SAP amendment is to follow the FDA comments:

FDA Response dated 28th March 2017 for type C meeting Question 7:

We agree that an asymptotic log-rank test instead of a permutation based log-rank test can be used as the primary analysis method. You may keep the permutation based logrank test as a secondary analysis method.

Another purpose is to revise the context to align with the amended protocol version 7.0 dated 13<sup>th</sup> July 2017. The following changes are made in this Statistical Analysis Plan (SAP) from the previous version of SAP due to the amendment to the protocol.

For primary endpoint, analysis method has changed to stratified log-rank test from the log-rank based permutation test.

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019

- Only treatment-emergent adverse events are collected in this study. Previously the SAP contained summaries of adverse events and treatment-emergent adverse events, the latter were removed to avoid redundancy.
- Detailed description on the identification of the following adverse event were added: serious infections, opportunistic infections, anaphylaxis, injection related reactions and injection site reactions.
- Detailed description of the following efficacy evaluation is added: EQ-5D Scoring and Visual acuity function.
- Detailed description of the immunogenicity and immunogenicity analyses were added.
- The analysis of relapse-free subjects using logistic regression will not be conducted because of a lot of early events.
- Clarify the definition of baseline ARR.
- Resolve inconsistencies mainly for scope of analysis in SAP.

#### 5.6 Amendment from Ver 6.0 to 6.1

The primary purpose of this SAP amendment is to update the amended protocol version 8.0 dated 18<sup>th</sup> June 2018.

### 5.7 Amendment from Ver 6.1 to 7.0

Related to: SOP-GDO-WW-019

The primary purpose of this SAP amendment is to include additional sensitivity analyses for the primary and key secondary endpoints:

- Sensitivity analysis for primary endpoint TFR (protocol-defined relapse) using stratified weighted log-rank test with Fleming-Harrington weight function was added.
- Sensitivity analysis for change from baseline in pain and fatigue was added, including additional information from the withdrawal and OLE baseline visits.
- Minor updates throughout the document to increase clarity and consistency.


#### REFERENCES

- [1] Rubin, DB. Multiple Imputation for Nonresponse in Surveys. New York: Wiley; 1987.
- [2] Little RJA. Missing-data adjustments in large surveys. J Buss Econ Stat. 1988; 6:287– 296.
- [3] Gold R, Kappos L, Arnold DL et al. Placebo-controlled phase 3 study of oral BG-12 for relapsing multiple sclerosis. N Engl J Med. 2012; 367: 1098-107.
- [4] Kappos L, Radue EW, O'Connor P et al. A placebo-controlled trial of oral fingolimod in relapsing multiple sclerosis. N Engl J Med. 2010; 362: 387-401.
- [5] Cree BA, Bennett JL, Sheehan M et al. Placebo-controlled study in neuromyelitis optica-Ethical and design considerations. Multi Scler 2015 published online.
- [6] Seung-Hwan Lee. On the versatility of the combination of the weighted log-rank statistic. Computational Statistics & Data Analysis. 2007; 51: 6557 - 6564

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019


#### **APPENDIX**

### 7.1 SAS code for primary and key secondary analysis

## Primary analysis for TFR

```
proc lifetest data = xxx;
class TREAT;
time TIME*CENS (1);
strata PRIORTHERAPY ATTACK / group = TREAT;
run;
```

#### Notation:

TREAT: treatment group (SA237 or Placebo),

TIME: time to first relapse. CENS: censoring variable,

PRIORTHERAPY: prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others),

ATTACK: the most recent attack in the last one year prior to screening (first attack or relapse).

## Sensitivity analysis for primary analysis

```
proc lifetest data = xxx;
class TREAT;
time TIME*CENS (1);
strata PRIORTHERAPY ATTACK / group = TREAT test=fleming(0,1);
run;
```

## Secondary analysis for pain and fatigue

```
proc mixed data = xxx;
 class TREAT;
 model CFBL = BL TREAT PRIORTHERAPY ATTACK;
Ismeans TREAT / pdiff cl
run;
```

## Notation:

TREAT: treatment group (SA237 or Placebo),

CFBL: change from baseline value of VAS or FACIT,

BL: baseline value of VAS or FACIT,

PRIORTHERAPY: prior therapy for prevention of NMO/NMOSD attack (B-cell depleting therapy or immunosuppressants/others),

ATTACK: the most recent attack in the last one year prior to screening (first attack or relapse)

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019

## 7.2 EQ-5D Scoring Algorithm:

This program computes the U.S. preference-weighted index score using self-reported EQ-5D data.

It is presumed that the data set includes the following 5 variables:

| Dimension | Variable Name | Range |
|--------------------|---------------|-------|
| Mobility | MO | 1-3 |
| Self-care | SC | 1-3 |
| Usual activities | UA | 1-3 |
| Pain/discomfort | PD | 1-3 |
| Anxiety/depression | AD | 1-3 |

Where a 1 indicates no problems, a 2 indicates moderate problems, and a 3 indicates severe problems.

To get U.S. EQ-5D index scores, paste data to the first 5 columns and read values from the last column.

The index score will not be generated when responses are missing for 1 or more of the 5 dimensions.

If there are more than 5,000 respondents, apply the algorithms for all the variables except the first 5 to more lines.

| МО | SC | UA | PD | AD | m1 | s1 | u1 | p1 | a1 | m2 | s2 | u2 | p2 | a2 | d1 | i2 | i22 | i3 | i32 | pred | full health | EQ-5D index(US_D1) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 0 | 0 | 4 | 16 | -0.1090707 | -0.109 | -0.1090707 |
| 3 | 3 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 4 | 0 | 0 | 3 | 9 | -0.0996728 | -0.100 | -0.0996728 |
| 3 | 3 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 3 | 9 | -0.0995382 | -0.100 | -0.0995382 |
| 3 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 4 | 0 | 0 | 3 | 9 | -0.0402381 | -0.040 | -0.0402381 |
| 3 | 2 | 3 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 4 | 0 | 0 | 3 | 9 | -0.0383556 | -0.038 | -0.0383556 |
| 3 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 3 | 9 | -0.02361 | -0.024 | -0.02361 |
| 3 | 3 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 1 | 1 | 2 | 4 | -0.0119344 | -0.012 | -0.0119344 |
| 3 | 2 | 2 | 3 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 1 | 1 | 2 | 4 | -0.0100519 | -0.010 | -0.0100519 |
| 3 | 1 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 3 | 9 | -0.002608 | -0.003 | -0.002608 |
| 3 | 3 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | -0.001113 | -0.001 | -0.001113 |
| 3 | 2 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.0007695 | 0.001 | 0.0007695 |
| 3 | 3 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 0.0153805 | 0.015 | 0.0153805 |
| 3 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 4 | 0.0155151 | 0.016 | 0.0155151 |


Related to: SOP-GDO-WW-019

| 3 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 3 | 9 | 0.0300077 | 0.030 | 0.0300077 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 | 1 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.0363825 | 0.036 | 0.0363825 |
| 3 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 4 | 0.0365171 | 0.037 | 0.0365171 |
| 3 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4 | 1 | 1 | 2 | 4 | 0.0493828 | 0.049 | 0.0493828 |
| 3 | 3 | 2 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1 | 1 | 2 | 4 | 0.0583114 | 0.058 | 0.0583114 |
| 3 | 3 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 3 | 9 | 0.0633035 | 0.063 | 0.0633035 |
| 3 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.0691328 | 0.069 | 0.0691328 |
| 3 | 2 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 0.0766977 | 0.077 | 0.0766977 |
| 2 | 3 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 0 | 0 | 3 | 9 | 0.0774663 | 0.077 | 0.0774663 |
| 1 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 3 | 9 | 0.0838874 | 0.084 | 0.0838874 |
| 3 | 2 | 2 | 3 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 4 | 1 | 1 | 0.0859055 | 0.086 | 0.0859055 |
| 3 | 1 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 0.0958172 | 0.096 | 0.0958172 |
| 3 | 3 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.102294 | 0.102 | 0.102294 |
| 3 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 0.1024286 | 0.102 | 0.1024286 |
| 2 | 3 | 2 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 1 | 1 | 2 | 4 | 0.10577 | 0.106 | 0.10577 |
| 3 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 4 | 0.1124453 | 0.112 | 0.1124453 |
| 2 | 3 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.1165914 | 0.117 | 0.1165914 |
| 3 | 3 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 4 | 1 | 1 | 2 | 4 | 0.1177461 | 0.118 | 0.1177461 |
| 3 | 2 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.1181005 | 0.118 | 0.1181005 |
| 3 | 2 | 3 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 2 | 4 | 0.1196286 | 0.120 | 0.1196286 |
| 1 | 3 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.1228779 | 0.123 | 0.1228779 |
| 1 | 3 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 4 | 0.1230125 | 0.123 | 0.1230125 |
| 3 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.134594 | 0.135 | 0.134594 |
| 3 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 4 | 0.145061 | 0.145 | 0.145061 |
| 3 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.1454154 | 0.145 | 0.1454154 |
| 3 | 1 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.1537135 | 0.154 | 0.1537135 |
| 3 | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 4 | 1 | 1 | 0.1542688 | 0.154 | 0.1542688 |
| 3 | 2 | 2 | 2 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 2 | 4 | 1 | 1 | 0.1561513 | 0.156 | 0.1561513 |
| 3 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 2 | 4 | 0.1617287 | 0.162 | 0.1617287 |
| 3 | 2 | 3 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.1636112 | 0.164 | 0.1636112 |
| 3 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.1645349 | 0.165 | 0.1645349 |
| 2 | 3 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 1 | 1 | 2 | 4 | 0.1652047 | 0.165 | 0.1652047 |
| 3 | 1 | 3 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.166063 | 0.166 | 0.166063 |


| 2 | 2 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 2 | 4 | 0.1670872 | 0.167 | 0.1670872 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 4 | 0.1783568 | 0.178 | 0.1783568 |
| 3 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.1810284 | 0.181 | 0.1810284 |
| 3 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0.181163 | 0.181 | 0.181163 |
| 1 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 0.1823126 | 0.182 | 0.1823126 |
| 1 | 2 | 3 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.1841951 | 0.184 | 0.1841951 |
| 3 | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.1864638 | 0.186 | 0.1864638 |
| 3 | 2 | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.1883463 | 0.188 | 0.1883463 |
| 2 | 3 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 0.1925196 | 0.193 | 0.1925196 |
| 1 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 4 | 0.1989407 | 0.199 | 0.1989407 |
| 3 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 0.1993588 | 0.199 | 0.1993588 |
| 2 | 3 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 2 | 4 | 1 | 1 | 0.2017274 | 0.202 | 0.2017274 |
| 3 | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2029573 | 0.203 | 0.2029573 |
| 2 | 2 | 2 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 4 | 1 | 1 | 0.2036099 | 0.204 | 0.2036099 |
| 2 | 1 | 3 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 2 | 4 | 0.2135216 | 0.214 | 0.2135216 |
| 3 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2137787 | 0.214 | 0.2137787 |
| 3 | 2 | 3 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 2 | 4 | 1 | 1 | 0.215586 | 0.216 | 0.215586 |
| 3 | 3 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.219625 | 0.220 | 0.219625 |
| 1 | 1 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 2 | 4 | 0.2199427 | 0.220 | 0.2199427 |
| 3 | 2 | 2 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.2215075 | 0.222 | 0.2215075 |
| 3 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.2239593 | 0.224 | 0.2239593 |
| 3 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2304464 | 0.230 | 0.2304464 |
| 3 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2323289 | 0.232 | 0.2323289 |
| 2 | 3 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2339224 | 0.234 | 0.2339224 |
| 3 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2347807 | 0.235 | 0.2347807 |
| 2 | 3 | 3 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 4 | 1 | 1 | 2 | 4 | 0.2354505 | 0.235 | 0.2354505 |
| 2 | 2 | 1 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0.2358049 | 0.236 | 0.2358049 |
| 1 | 3 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2402089 | 0.240 | 0.2402089 |
| 1 | 2 | 2 | 3 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0.2420914 | 0.242 | 0.2420914 |
| 3 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2469399 | 0.247 | 0.2469399 |
| 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0.2470745 | 0.247 | 0.2470745 |
| 2 | 3 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2504159 | 0.250 | 0.2504159 |
| 1 | 3 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2510303 | 0.251 | 0.2510303 |


| 1 | 3 | 3 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.2525584 | 0.253 | 0.2525584 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | 2 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2529128 | 0.253 | 0.2529128 |
| 3 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 3 | 9 | 0 | 0 | 0.2603277 | 0.260 | 0.2603277 |
| 2 | 3 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2612373 | 0.261 | 0.2612373 |
| 2 | 2 | 3 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 2 | 4 | 1 | 1 | 0.2630446 | 0.263 | 0.2630446 |
| 3 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2642745 | 0.264 | 0.2642745 |
| 1 | 3 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.2675238 | 0.268 | 0.2675238 |
| 1 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0.2676584 | 0.268 | 0.2676584 |
| 3 | 1 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2679419 | 0.268 | 0.2679419 |
| 3 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0.2680765 | 0.268 | 0.2680765 |
| 2 | 1 | 2 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 0.2714179 | 0.271 | 0.2714179 |
| 2 | 3 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 2 | 4 | 1 | 1 | 0.2719732 | 0.272 | 0.2719732 |
| 2 | 3 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 4 | 0.2794331 | 0.279 | 0.2794331 |
| 3 | 2 | 3 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.2809422 | 0.281 | 0.2809422 |
| 2 | 1 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2822393 | 0.282 | 0.2822393 |
| 3 | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.283394 | 0.283 | 0.283394 |
| 1 | 3 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 0.2858542 | 0.286 | 0.2858542 |
| 1 | 1 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0.2885258 | 0.289 | 0.2885258 |
| 1 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0.2886604 | 0.289 | 0.2886604 |
| 1 | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3015261 | 0.302 | 0.3015261 |
| 2 | 3 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.3041682 | 0.304 | 0.3041682 |
| 2 | 2 | 2 | 3 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 3 | 9 | 0 | 0 | 0.3077863 | 0.308 | 0.3077863 |
| 3 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3082571 | 0.308 | 0.3082571 |
| 1 | 3 | 2 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.3104547 | 0.310 | 0.3104547 |
| 3 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3107089 | 0.311 | 0.3107089 |
| 2 | 2 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3117331 | 0.312 | 0.3117331 |
| 3 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3138963 | 0.314 | 0.3138963 |
| 1 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.3212761 | 0.321 | 0.3212761 |
| 3 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3273766 | 0.327 | 0.3273766 |
| 1 | 2 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.328841 | 0.329 | 0.328841 |
| 3 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3303898 | 0.330 | 0.3303898 |
| 2 | 1 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3308526 | 0.331 | 0.3308526 |
| 2 | 3 | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 4 | 2 | 4 | 1 | 1 | 0.3314079 | 0.331 | 0.3314079 |


| Ī | 2 | 2 | 3 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 2 | 4 | 1 | 1 | 0.3332904 | 0.333 | 0.3332904 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 2 | 3 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.3373294 | 0.337 | 0.3373294 |
| | 3 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0.3440047 | 0.344 | 0.3440047 |
| | 3 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3470575 | 0.347 | 0.3470575 |
| | 1 | 1 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3479605 | 0.348 | 0.3479605 |
| | 2 | 3 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.3481508 | 0.348 | 0.3481508 |
| | 3 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3495093 | 0.350 | 0.3495093 |
| | 1 | 3 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.3544373 | 0.354 | 0.3544373 |
| | 1 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0.3545719 | 0.355 | 0.3545719 |
| | 2 | 1 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3581675 | 0.358 | 0.3581675 |
| | 2 | 2 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3613549 | 0.361 | 0.3613549 |
| | 3 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.3625848 | 0.363 | 0.3625848 |
| | 1 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0.3645886 | 0.365 | 0.3645886 |
| | 1 | 2 | 2 | 3 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3676414 | 0.368 | 0.3676414 |
| | 1 | 3 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3698894 | 0.370 | 0.3698894 |
| | 1 | 2 | 3 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.3717719 | 0.372 | 0.3717719 |
| | 2 | 3 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 3 | 9 | 0 | 0 | 0.3761496 | 0.376 | 0.3761496 |
| | 2 | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3778484 | 0.378 | 0.3778484 |
| | 2 | 2 | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 9 | 0 | 0 | 0.3780321 | 0.378 | 0.3780321 |
| | 3 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.3792525 | 0.379 | 0.3792525 |
| | 2 | 3 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3800964 | 0.380 | 0.3800964 |
| | 3 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.3817043 | 0.382 | 0.3817043 |
| | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.395746 | 0.396 | 0.395746 |
| | 2 | 3 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 1 | 0.3967641 | 0.397 | 0.3967641 |
| | 2 | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 4 | 0 | 0 | 0.3969679 | 0.397 | 0.3969679 |
| | 1 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.3972043 | 0.397 | 0.3972043 |
| | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.3981978 | 0.398 | 0.3981978 |
| | 2 | 2 | 3 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.3986466 | 0.399 | 0.3986466 |
| | 1 | 2 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.3998364 | 0.400 | 0.3998364 |
| | 2 | 1 | 3 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 1 | 0.4010984 | 0.401 | 0.4010984 |
| | 3 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4065674 | 0.407 | 0.4065674 |
| J | 3 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4090192 | 0.409 | 0.4090192 |
| | 2 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4100434 | 0.410 | 0.4100434 |


| | 1 | 3 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.413872 | 0.414 | 0.413872 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 3 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4148655 | 0.415 | 0.4148655 |
| | 1 | 2 | 3 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.4157545 | 0.416 | 0.4157545 |
| | 1 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4163299 | 0.416 | 0.4163299 |
| | 1 | 1 | 3 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.4182063 | 0.418 | 0.4182063 |
| | 2 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0.424079 | 0.424 | 0.424079 |
| | 3 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4256869 | 0.426 | 0.4256869 |
| | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4271513 | 0.427 | 0.4271513 |
| | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4291629 | 0.429 | 0.4291629 |
| | 2 | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.4297182 | 0.430 | 0.4297182 |
| | 1 | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0.4305001 | 0.431 | 0.4305001 |
| | 2 | 2 | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 0.4316007 | 0.432 | 0.4316007 |
| | 1 | 1 | 2 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4354494 | 0.435 | 0.4354494 |
| | 1 | 3 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.4360047 | 0.436 | 0.4360047 |
| | 2 | 2 | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 3 | 9 | 0 | 0 | 0.4374668 | 0.437 | 0.4374668 |
| | 1 | 2 | 2 | 2 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 0.4378872 | 0.438 | 0.4378872 |
| | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4421804 | 0.442 | 0.4421804 |
| | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.442315 | 0.442 | 0.442315 |
| | 2 | 1 | 3 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0.445081 | 0.445 | 0.445081 |
| | 2 | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4456564 | 0.446 | 0.4456564 |
| | 2 | 3 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.4462117 | 0.446 | 0.4462117 |
| | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4462708 | 0.446 | 0.4462708 |
| | 1 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0.4515021 | 0.452 | 0.4515021 |
| | 2 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4564778 | 0.456 | 0.4564778 |
| | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4627643 | 0.463 | 0.4627643 |
| | 2 | 3 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.4628794 | 0.463 | 0.4628794 |
| | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0.4628989 | 0.463 | 0.4628989 |
| | 2 | 2 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 0.4647619 | 0.465 | 0.4647619 |
| | 2 | 1 | 2 | 2 | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 0 | 0 | 0.4672137 | 0.467 | 0.4672137 |
| | 1 | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4681997 | 0.468 | 0.4681997 |
| J | 1 | 2 | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.4700822 | 0.470 | 0.4700822 |
| | 2 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4784067 | 0.478 | 0.4784067 |
| | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4846932 | 0.485 | 0.4846932 |


| | 2 | 3 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.4950744 | 0.495 | 0.4950744 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.4955146 | 0.496 | 0.4955146 |
| | 2 | 2 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.4969569 | 0.497 | 0.4969569 |
| | 1 | 2 | 3 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.4973219 | 0.497 | 0.4973219 |
| | 2 | 1 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.4994087 | 0.499 | 0.4994087 |
| | 1 | 3 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5013609 | 0.501 | 0.5013609 |
| | 1 | 2 | 2 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.5032434 | 0.503 | 0.5032434 |
| | 1 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.5056952 | 0.506 | 0.5056952 |
| | 2 | 2 | 3 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.5075289 | 0.508 | 0.5075289 |
| | 2 | 3 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5115679 | 0.512 | 0.5115679 |
| | 1 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.5121823 | 0.512 | 0.5121823 |
| | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0.5140648 | 0.514 | 0.5140648 |
| | 1 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0.5165166 | 0.517 | 0.5165166 |
| | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.5223893 | 0.522 | 0.5223893 |
| | 2 | 2 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.5241966 | 0.524 | 0.5241966 |
| | 2 | 1 | 3 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 0 | 0 | 0.5266484 | 0.527 | 0.5266484 |
| | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.5286758 | 0.529 | 0.5286758 |
| | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.5288104 | 0.529 | 0.5288104 |
| | 2 | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0.5325699 | 0.533 | 0.5325699 |
| | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0.5433913 | 0.543 | 0.5433913 |
| | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5460104 | 0.546 | 0.5460104 |
| | 1 | 1 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0.5496778 | 0.550 | 0.5496778 |
| | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0.5498124 | 0.550 | 0.5498124 |
| | 1 | 2 | 3 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5626781 | 0.563 | 0.5626781 |
| | 1 | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5651299 | 0.565 | 0.5651299 |
| | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5728851 | 0.573 | 0.5728851 |
| | 2 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5753369 | 0.575 | 0.5753369 |
| | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.589993 | 0.590 | 0.589993 |
| | 2 | 1 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0.5920046 | 0.592 | 0.5920046 |
| | 1 | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.5924448 | 0.592 | 0.5924448 |
| | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 16 | 0 | 0 | 0.5971891 | 0.597 | 0.5971891 |
| | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.6091125 | 0.609 | 0.6091125 |
| 1 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0.6193195 | 0.619 | 0.6193195 |


| 1 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.6257406 | 0.626 | 0.6257406 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 2 | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 0 | 0 | 0.6721313 | 0.672 | 0.6721313 |
| 1 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 0 | 0 | 0.6784178 | 0.678 | 0.6784178 |
| 2 | 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 0 | 0 | 0.6886248 | 0.689 | 0.6886248 |
| 2 | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 0 | 0 | 0.7052925 | 0.705 | 0.7052925 |
| 2 | 1 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 9 | 0 | 0 | 0.7077443 | 0.708 | 0.7077443 |
| 1 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7319864 | 0.732 | 0.7319864 |
| 2 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7421934 | 0.742 | 0.7421934 |
| 1 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7484799 | 0.748 | 0.7484799 |
| 2 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7588611 | 0.759 | 0.7588611 |
| 2 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7613129 | 0.761 | 0.7613129 |
| 1 | 2 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7651476 | 0.765 | 0.7651476 |
| 1 | 1 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7675994 | 0.768 | 0.7675994 |
| 2 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7753546 | 0.775 | 0.7753546 |
| 2 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7778064 | 0.778 | 0.7778064 |
| 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.7806749 | 0.781 | 0.7806749 |
| 2 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 0 | 0.7944741 | 0.794 | 0.7944741 |
| 1 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.7973426 | 0.797 | 0.7973426 |
| 1 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.7997944 | 0.800 | 0.7997944 |
| 2 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8075496 | 0.808 | 0.8075496 |
| 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8100014 | 0.810 | 0.8100014 |
| 1 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8138361 | 0.814 | 0.8138361 |
| 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8162879 | 0.816 | 0.8162879 |
| 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.8246575 | 0.825 | 0.8246575 |
| 2 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8266691 | 0.827 | 0.8266691 |
| 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.8271093 | 0.827 | 0.8271093 |
| 1 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8329556 | 0.833 | 0.8329556 |
| 2 | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0.8431626 | 0.843 | 0.8431626 |
| 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.843777 | 0.844 | 0.843777 |
| 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.853984 | 0.854 | 0.853984 |
| 1 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0.8602705 | 0.860 | 0.8602705 |
| 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | -1 | 0 | 0 | 0 | 0 | 0.8604051 | 1.000 | 1 |


## 7.3 Procedure to identify the clinical relapse of optic neuritis occurred in the doubleblind period:

The clinical relapse of optic neuritis occurred in the double-blind period of SA-309JG study will be identified by satisfying with either or both of followings. The Relapse Assessment Form (RAF) completed by study sites will be used for the identification.

- Lower box "New or worsening neurological symptoms relating to this functional area reported by the patient at this visit. Please describe:" is ticked in the Section A-1 "Visual (optic) functions: Symptoms" of the RAF, and then the information is described per the instruction.
- The information on new or worsening neurological symptoms in visual (optic) functions are described in section B of RAF.

## [Reference: Section A-1 of RAF]

| 1. V | isual(optic)functions. |
|---|---|
| > | Symptoms. |
| | No new or worsening neurological symptoms in this functional area from the previous assessment of EDSS/FSS. |
| | New or worsening neurological symptoms relating to this functional area reported by the patient at this visit. Please describe: |

TP-GDO-WW-016-01 Confidential Version 7.0 Version Date: 28NOV2018 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019


# 7.4 MedDRA basket

# Opportunistic infections

| Opportumstic i | in cenons | | | | |
|---|---|---|---|---|---|
| Meningomyelitis<br>herpes | Capnocytophaga test positive | Eye infection toxoplasmal | Histoplasmosis<br>disseminated | Mycobacterium ulcerans infection | Pulmonary<br>trichosporonosis |
| Abscess fungal | Central nervous<br>system fungal<br>infection | Eye infection viral | Human<br>anaplasmosis | Mycotic corneal ulcer | Pulmonary<br>tuberculoma |
| Acid fast bacilli infection | Central nervous<br>system viral<br>infection | Female genital tract tuberculosis | Human<br>bocavirus<br>infection | Mycotic endophthalmitis | Pulmonary<br>tuberculosis |
| Acinetobacter bacteraemia | Cerebral aspergillosis | Flavobacterium infection | Human ehrlichiosis | Myocarditis mycotic | Pyelonephritis<br>fungal |
| Acinetobacter infection | Cerebral candidiasis | Focal epithelial hyperplasia | Human<br>herpesvirus 8<br>infection | Myocarditis<br>toxoplasmal | Q fever |
| Acute haemorrhagic conjunctivitis | Cerebral fungal infection | Fungaemia | Indeterminate<br>leprosy | Nasal herpes | Raoultella ornithinolytica infection |
| Acute hepatitis B | Cerebral<br>toxoplasmosis | Fungal abscess<br>central nervous<br>system | Infection in an immunocompro mised host | Necrotising fasciitis fungal | Renal<br>tuberculosis |
| Acute hepatitis C | Cervix warts | Fungal cystitis | Intestinal<br>tuberculosis | Necrotising<br>herpetic<br>retinopathy | Respiratory moniliasis |
| Acute pulmonary histoplasmosis | Chromoblastomy cosis | Fungal endocarditis | Isosporiasis | Neurocryptococc osis | Respiratory tract infection fungal |
| Adrenal gland tuberculosis | Chronic<br>pulmonary<br>histoplasmosis | Fungal<br>labyrinthitis | JC virus granule cell neuronopathy | Neutropenic infection | Retinitis<br>histoplasma |
| Aeromonas infection | Coccidioides encephalitis | Fungal<br>oesophagitis | JC virus infection | Neutropenic sepsis | Retinitis viral |
| Aeromonas test positive | Coccidioidomyc osis | Fungal peritonitis | JC virus test | Nocardia sepsis | Rhodococcus infection |
| Alcaligenes infection | Colitis herpes | Fungal<br>pharyngitis | JC virus test positive | Nocardia test positive | Rhodococcus<br>test positive |
| Allescheriosis | Conjunctivitis tuberculous | Fungal retinitis | Joint tuberculosis | Nocardiosis | Salpingitis<br>tuberculous |
| Alternaria infection | Coxiella infection | Fungal sepsis | Kaposi's sarcoma | Oesophageal candidiasis | Scedosporium infection |
| Amoebiasis | Creutzfeldt-<br>Jakob disease | Fungal tracheitis | Kaposi's sarcoma<br>AIDS related | Oesophageal<br>tuberculosis | Sepsis<br>pasteurella |
| Amoebic brain abscess | Cronobacter infection | Fusarium infection | Kaposi's<br>varicelliform<br>eruption | Ophthalmic<br>herpes simplex | Shewanella algae<br>bacteraemia |
| Amoebic colitis | Cronobacter<br>necrotising<br>enterocolitis | Gastritis fungal | Keratitis fungal | Ophthalmic<br>herpes zoster | Sinusitis<br>aspergillus |

TP-GDO-WW-016-01 Effective Date: 28Aug13 Related to: SOP-GDO-WW-019 Confidential


| Amoebic dysentery | Cryptococcal cutaneous infection | Gastritis herpes | Keratitis viral | Opportunistic infection | Sinusitis fungal |
|---|---|---|---|---|---|
| Amoebic lung abscess | Cryptococcal fungaemia | Gastroenteritis cryptococcal | Keratouveitis | Oral candidiasis | Sphingomonas<br>paucimobilis<br>infection |
| Amoebic skin<br>ulcer | Cryptococcosis | Gastroenteritis cryptosporidial | Laryngitis fungal | Oral fungal infection | Spleen<br>tuberculosis |
| Anal fungal infection | Cryptococcus<br>test | Gastrointestinal candidiasis | Legionella infection | Oral hairy<br>leukoplakia | Splenic candidiasis |
| Angina gangrenous | Cryptococcus test positive | Gastrointestinal fungal infection | Lepromatous leprosy | Oral herpes | Splenic infection fungal |
| Angiostrongylus infection | Cryptosporidiosi s infection | Genital herpes | Leprosy | Oral tuberculosis | Stenotrophomon as infection |
| Anogenital warts | Cutaneous<br>coccidioidomyco<br>sis | Genital herpes simplex | Leptotrichia infection | Oro-pharyngeal aspergillosis | Stenotrophomon as sepsis |
| Anorectal human papilloma virus infection | Cutaneous<br>tuberculosis | Genital herpes zoster | Leuconostoc infection | Oropharyngeal candidiasis | Stomatococcal infection |
| Anti-JC virus antibody index | Cytomegalovirus chorioretinitis | Granulicatella bacteraemia | Listeria<br>encephalitis | Oropharyngitis<br>fungal | Stomatococcus test positive |
| Arthritis fungal | Cytomegalovirus colitis | Granulicatella infection | Listeria sepsis | Orthopox virus infection | Strongyloidiasis |
| Aspergilloma | Cytomegalovirus duodenitis | Hepatic candidiasis | Listeria test positive | Osteomyelitis<br>blastomyces | Superinfection fungal |
| Aspergillosis oral | Cytomegalovirus enteritis | Hepatic infection fungal | Listeriosis | Osteomyelitis fungal | Superinfection mycobacterial |
| Aspergillus infection | Cytomegalovirus enterocolitis | Hepatitis B | Lower<br>respiratory tract<br>herpes infection | Otitis media<br>fungal | Systemic candida |
| Aspergillus test | Cytomegalovirus<br>gastritis | Hepatitis C | Lower respiratory tract infection fungal | Pancreatitis<br>fungal | Systemic<br>mycosis |
| Aspergillus test positive | Cytomegalovirus gastroenteritis | Hepatitis<br>toxoplasmal | Lower respiratory tract infection viral | Pantoea<br>agglomerans<br>infection | Thyroid<br>tuberculosis |
| Atypical<br>mycobacterial<br>infection | Cytomegalovirus<br>gastrointestinal<br>infection | Hepatosplenic candidiasis | Lupus vulgaris | Paracoccidioides infection | Tonsillitis fungal |
| Atypical<br>mycobacterial<br>lower respiratory<br>tract infection | Cytomegalovirus<br>gastrointestinal<br>ulcer | Herpes<br>oesophagitis | Lymph node tuberculosis | Parasitic<br>encephalitis | Toxoplasmosis |
| Atypical<br>mycobacterial<br>lymphadenitis | Cytomegalovirus<br>hepatitis | Herpes<br>ophthalmic | Lymphadenitis<br>fungal | Parvimonas<br>infection | Tuberculoid<br>leprosy |
| Atypical<br>mycobacterial<br>pneumonia | Cytomegalovirus infection | Herpes<br>pharyngitis | Male genital tract tuberculosis | Parvimonas<br>micra infection | Tuberculoma of<br>central nervous<br>system |


| Atypical<br>mycobacterium<br>pericarditis | Cytomegalovirus<br>mucocutaneous<br>ulcer | Herpes sepsis | Meningitis<br>aspergillus | | |
|---|---|---|---|---|---|
| Atypical pneumonia | Cytomegalovirus<br>myelomeningora<br>diculitis | Herpes simplex | Meningitis<br>candida | Penicillium infection | Tuberculosis<br>bladder |
| Babesiosis | Cytomegalovirus<br>myocarditis | Herpes simplex cervicitis | Meningitis coccidioides | Pericarditis<br>fungal | Tuberculosis gastrointestinal |
| Bacillary angiomatosis | Cytomegalovirus oesophagitis | Herpes simplex colitis | Meningitis cronobacter | Pericarditis<br>histoplasma | Tuberculosis<br>liver |
| Balamuthia infection | Cytomegalovirus pancreatitis | Herpes simplex encephalitis | Meningitis cryptococcal | Pericarditis<br>tuberculous | Tuberculosis of central nervous system |
| BK virus infection | Cytomegalovirus pericarditis | Herpes simplex gastritis | Meningitis<br>exserohilum | Peritoneal candidiasis | Tuberculosis of eye |
| Blastocystis infection | Cytomegalovirus syndrome | Herpes simplex hepatitis | Meningitis<br>fungal | Peritoneal tuberculosis | Tuberculosis of genitourinary system |
| Blastomycosis | Cytomegalovirus<br>test | Herpes simplex meningitis | Meningitis<br>herpes | Phaehyphomyco sis | Tuberculosis of intrathoracic lymph nodes |
| Bone<br>tuberculosis | Cytomegalovirus test positive | Herpes simplex<br>meningoencepha<br>litis | Meningitis<br>histoplasma | Pharyngeal<br>abscess | Tuberculosis of peripheral lymph nodes |
| Borderline<br>leprosy | Cytomegalovirus<br>urinary tract<br>infection | Herpes simplex meningomyelitis | Meningitis<br>listeria | Pneumocystis<br>jirovecii<br>infection | Tuberculosis<br>ureter |
| Botryomycosis | Cytomegalovirus<br>viraemia | Herpes simplex necrotising retinopathy | Meningitis<br>toxoplasmal | Pneumocystis<br>jirovecii<br>pneumonia | Tuberculous<br>abscess central<br>nervous system |
| Bovine<br>tuberculosis | Dengue fever | Herpes simplex oesophagitis | Meningitis<br>tuberculous | Pneumocystis test positive | Tuberculous endometritis |
| Brachyspira infection | Disseminated Bacillus Calmette-Guerin infection | Herpes simplex otitis externa | Meningoencepha<br>litis herpes<br>simplex neonatal | Pneumonia<br>blastomyces | Tuberculous<br>laryngitis |
| Brevibacterium infection | Disseminated cryptococcosis | Herpes simplex pharyngitis | Meningoencepha<br>litis herpetic | Pneumonia<br>cryptococcal | Tuberculous pleurisy |
| Bronchitis fungal | Disseminated cytomegaloviral infection | Herpes simplex pneumonia | Meningoencepha<br>litis viral | Pneumonia<br>cytomegaloviral | Tuberculous tenosynovitis |
| Bronchopulmona ry aspergillosis | Disseminated tuberculosis | Herpes simplex sepsis | Methylobacteriu<br>m infection | Pneumonia<br>fungal | Upper<br>respiratory<br>fungal infection |
| Burkholderia<br>cepacia complex<br>infection | Disseminated<br>varicella zoster<br>vaccine virus<br>infection | Herpes simplex visceral | Microsporidia infection | Pneumonia<br>herpes viral | Urinary tract infection fungal |


| Burkholderia<br>cepacia complex<br>sepsis | Ear tuberculosis | Herpes virus infection | Miliary Pneumonia pneumonia legionella | | Variant<br>Creutzfeldt-<br>Jakob disease |
|---|---|---|---|---|---|
| Burkholderia gladioli infection | Encephalitis cytomegalovirus | Herpes zoster | Mucocutaneous candidiasis | Pneumonia<br>toxoplasmal | Varicella |
| Burkholderia<br>infection | Encephalitis<br>fungal | Herpes zoster<br>cutaneous<br>disseminated | Mucormycosis | Polyomavirus-<br>associated<br>nephropathy | Varicella<br>keratitis |
| Burkholderia<br>mallei infection | Encephalitis post<br>varicella | Herpes zoster disseminated | Mycetoma<br>mycotic | Porphyromonas infection | Varicella zoster gastritis |
| Burkholderia<br>pseudomallei<br>infection | Endocarditis<br>candida | Herpes zoster<br>infection<br>neurological | Mycobacterial infection | Presumed ocular<br>histoplasmosis<br>syndrome | Varicella zoster oesophagitis |
| Burkholderia test positive | Endocarditis<br>histoplasma | Herpes zoster<br>meningitis | Mycobacterial peritonitis | Progressive<br>multifocal<br>leukoencephalop<br>athy | Varicella zoster pneumonia |
| Candida endophthalmitis | Endocarditis Q<br>fever | Herpes zoster<br>meningoencepha<br>litis | Mycobacterium<br>abscessus<br>infection | Progressive vaccinia | Varicella zoster virus infection |
| Candida infection | Enterocolitis<br>fungal | Herpes zoster<br>meningomyelitis | Mycobacterium<br>avium complex<br>immune<br>restoration<br>disease | Prostatitis<br>tuberculous | Viral<br>keratouveitis |
| Candida<br>osteomyelitis | Epididymitis<br>blastomyces | Herpes zoster<br>necrotising<br>retinopathy | Mycobacterium<br>avium complex<br>infection | Pseudallescheria infection | Viral myelitis |
| Candida pneumonia | Epididymitis<br>tuberculous | Herpes zoster oticus | Mycobacterium chelonae infection | Pseudallescheria<br>sepsis | Viral<br>oesophagitis |
| Candida retinitis | Exserohilum infection | Herpes zoster pharyngitis | Mycobacterium<br>fortuitum<br>infection | Pseudomonal sepsis | Viral sepsis |
| Candida sepsis | Extrapulmonary tuberculosis | Histoplasmosis | Mycobacterium<br>kansasii<br>infection | Pseudomonas<br>aeruginosa<br>meningitis | Viral uveitis |
| Capnocytophaga infection | Eye infection fungal | Histoplasmosis cutaneous | Mycobacterium marinum infection | Pulmonary<br>mycosis | Yersinia sepsis |

# 7.5 Laboratory Data Conversion and Transformation Rules

• Conversion to Système International (SI) Units

Laboratory data should be stored on the database in the units in which they were originally delivered by the laboratory.

For analysis and reporting purposes, the data will be converted to SI units to allow the comparison of data delivered in different original units.

Results that include inequality sign will be converted into a numeric form removing inequality sign.

TP-GDO-WW-016-01 Confidential Version 7.0 Effective Date: 28Aug13 Version Date: 28NOV2018 Related to: SOP-GDO-WW-019


Results that cannot be converted into an expected numeric form nor interpreted, such as alphabetic entries like "adequate", will usually not be further processed, but displayed in patient listings.

### Marked Laboratory Abnormalities

For each laboratory test, a Marked Abnormality Range has been defined. A value outside of this range is considered to be potentially clinically relevant. This Marked Abnormality Range is wider than the Reference Range.

In addition, for each laboratory test, a percentage change, as an increase and/or decrease, has been defined which represents a clinically relevant change from baseline.

A Marked Abnormality is therefore defined as a test result:

which is outside of the Marked Abnormality Range, and which also represents a clinically relevant change from baseline of at least the designated amount during or within 30 days after end of trial treatment.

Baseline is taken as the last valid value before starting treatment. If no baseline is available, the midpoint of the Reference Range will be substituted for processing purposes for determination of Marked Abnormalities.

For urinalysis a missing baseline value will be replaced by 0 (zero).

NOTE: For calculating means and mean changes over time, missing values will not be included. If no baseline is available, no change from baseline will be calculated.

Values above and below the Reference Range are flagged on the listing by H and L. respectively. Marked Abnormalities are flagged by HH or LL.

Reference Ranges

Related to: SOP-GDO-WW-019


| Laboratory<br>Test Class | Laboratory Test | SI Unit | Reference Range [1,2] | Marked<br>Abnormality<br>Range | Direction of<br>Change | Relevant<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| Hematology | Hematocrit | fraction | M: 0.37 – 0.49<br>F: 0.36 – 0.46 b | 0.31 - 0.56 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| | Hemoglobin | g/L | M: 130 – 180<br>F: 120 – 160 b | 110-200 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| | Leukocytes (WBC) | 10°/L | 4.5 – 11.0 | 3.0 - 18.0 | Increase<br>Decrease | ≥ 30%<br>≥ 30% |
| | Platelets | 10 <sup>9</sup> /L | 150 - 350 | 100 - 550 | Increase<br>Decrease | ≥ 50%<br>≥ 30% |
| | Mean corpuscular<br>hemoglobin (MCH) | pg/cell | 25.0 - 35.0 | 21.2 - 40.2 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| | Mean corpuscular<br>hemoglobin concentration<br>(MCHC) | g/L | 310 – 370 | 260 – 430 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| | Mean corpuscular volume<br>(MCV) | tl. | 78 – 100 | 66 - 115 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| | Erythrocytes (RBC) | 10 <sup>12</sup> /L | M: 4.50 – 5.30<br>F: 4.10 – 5.10 b | 3.80 - 6.10 | Increase<br>Decrease | ≥ 15%<br>≥ 15% |
| Differentials | Bands | 109/L | 0-0.70 | 0-1.40 | Increase | ≥ 30% |
| | Bands | fraction | 0 - 0.05 | 0 - 0.10 | Increase | ≥ 30% |
| | Basophils | 109/L | 0-0.20 | 0 - 0.40 | Increase | ≥ 100% |
| | Basophils | fraction | 0-0.03 | 0 - 0.06 | Increase | ≥ 100% |
| | Lymphocytes | 10°/L | 1.00 - 4.80 | 0.70 - 7.60 | Increase<br>Decrease | ≥ 30%<br>≥ 30% |
| | Lymphocytes | fraction | 0.16 - 0.46 | 0.10 - 0.72 | Increase<br>Decrease | ≥ 30%<br>≥ 30% |
| | Monocytes | 109/L | 0 - 0.80 | 0 - 1.70 | Increase | ≥ 100% |
| | Monocytes | fraction | 0-0.11 | 0-0.22 | Increase | ≥ 100% |
| | Neutrophils | 10 <sup>9</sup> /L | 1.80 - 7.70 | 1.50 - 9.25 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | Neutrophils | fraction | 0.45 - 0.75 | 0.37 - 0.90 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | Eosinophils | 10°/L | 0-0.45 | 0-0.90 | Increase | ≥ 100% |
| | Eosinophils | fraction | 0 - 0.08 | 0-0.16 | Increase | ≥ 100% |
| Coagulation | Prothrombin Time,<br>normalized ratio (PTINR) | ratio | 0.70 - 1.30 | ≤ 2.00 | Increase | ≥ 30% |
| | Partial Thromboplastin<br>Time, activated (PTT) | seconds | 22.1 - 34.1 | 0-45 | Increase | ≥ 40% |
| | Fibrinogen | g/L | 1.75 - 4.00 a | ≥ 1.30 | Decrease | ≥30% |
| | Antithrombin 3 | fraction | 0.80 - 1.30 | ≥ 0.60 | Decrease | ≥ 20% |
| Heart Function | ASAT (SGOT) | U/L | M: 0-40°<br>F: 0-25 <sup>b</sup> | 0-80 | Increase | ≥ 50% |
| | Lactic Dehydrogenase<br>(LDH) | U/L | 0-210° | 0-420 | Increase | ≥ 50% |
| | Creatine phosphokinase<br>(CPK) total | U/L | M: 60 – 400 <sup>a</sup><br>F: 40 – 150 <sup>b</sup> | ≤ 800 | Increase | ≥ 50% |
| | CPK (MB Fraction) | μg/L | 0-5° | < 5 | Increase | 0% |

| Laboratory<br>Test Class | Laboratory Test | SI Unit | Reference Range [1,2] | Marked<br>Abnormality<br>Range | Direction of<br>Change | Clinically<br>Relevant<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|
| Liver Function | Alkaline Phosphatase | U/L | M: 0 - 115°<br>F: 0 - 100° | 0-220 | Increase | ≥ 50% |
| | ALAT (SGPT) | U/L | M: 0-55°<br>F: 0-30° | 0-110 | Increase | ≥ 50% |
| | Total Bilirubin | μmol/L | 0-17° | 0-34 | Increase | ≥ 75% |
| | Direct bilirubin | μmol/L | 0-7° | 0-14 | Increase | ≥ 75% |
| | γ-GTP | U/L | M: 0 - 94°<br>F: 0 - 70° | 0-190 | Increase | ≥ 50% |
| Renal Function | BUN | mmol/L | 2.9 - 8.9 | 0 - 14.3 | Increase | ≥ 50% |
| | Creatinine | μmol/L | 0-133 | 0-154 | Increase | ≥ 50% |
| Thyroid | Triiodothyronine (T3) | nmol/L | 0.92 - 2.78 | 0.74 - 3.30 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| Function | Thyroxine (T4) | nmol/L | 58 - 140 | 30 - 164 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | Free T4 | pmol/L | 10 – 36 | 5-40 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | TSH | mU/L | 0-5.0° | 0-10.0 | Increase | ≥ 30% |
| Protein | Albumin | g/L | 35.0 - 55.0 | ≥ 30 | Decrease | ≥ 20% |
| | Total Protein | g/L | 60 - 80 | 55 - 87 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| Lipid | Triglycerides (fasting) | mmol/L | 0.45 - 1.69 | 0-2.83 | Increase | ≥ 100% |
| Chemistry | Cholesterol | mmol/L | 0-6.18 | 0-8.30 | Increase | ≥ 30% |
| | LDL-Cholesterol | mmol/L | 0-4.13 | 0-5.4 | Increase | ≥ 30% |
| | HDL-Cholesterol | mmol/L | ≥ 0.91 | ≥ 0.65 | Decrease | ≥ 30% |
| Electrolytes | Chloride | mmol/L | 100 - 108 | 95 – 115 | Increase<br>Decrease | ≥ 7%<br>≥ 7% |
| | Potassium | mmol/L | 3.4-4.8 | 2.9 – 5.8 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | Sodium | mmol/L | 135 – 145 | 130-150 | Increase<br>Decrease | ≥ 7%<br>≥ 7% |
| | Bicarbonate | mmol/L | 22 – 26 | 18 – 28 | Increase<br>Decrease | ≥ 20%<br>≥ 20% |
| | Calcium | mmol/L | 2.10 - 2.60 | 2.00 - 2.90 | Increase<br>Decrease | ≥ 10%<br>≥ 10% |
| | Phosphorus inorganic | mmol/L | 0.84 - 1.45 | 0.75 - 1.60 | Increase<br>Decrease | ≥ 30%<br>≥ 30% |
| | Blood Glucose (fasting) | mmol/L | 3.90 - 6.10 | 2.80 - 11.10 | Increase<br>Decrease | ≥ 75%<br>≥ 75% |
| | Uric Acid | μmol/L | M: 214 – 506<br>F: 137 – 393 b | 0-600 | Increase | ≥ 50% |
| Urinalysis | Proteinuria | 1 to 6 | 1-3 | 1-3 | Increase | $\geq 2$ units <sup>d</sup> |
| Dipstick | Glycosuria | 1 to 6 | 1-3 | 1-3 | Increase | $\geq 2$ units d |
| | Hematuria | 1 to 6 | 1-3 | 1 – 3 | Increase | $\geq 2$ units d |
| | Leukocyturia | 1 to 6 | 1-3 | 1-3 | Increase | $\geq 2$ units d |
| Urinalysis | Casts | /HPF | 0-2 | 0-2 | Increase | ≥ 2 units |
| Microscopic e | WBCs | /HPF | 0-2 | 0-2 | Increase | ≥ 2 units |
| | RBCs | /HPF | 0-2 | 0-2 | Increase | ≥ 2 units |
| | Urinary spec. gravity f | No unit | 1.001 - 1.035 | not defined | not defined | not defined |

- a) For reporting and analyzing, the data are linearly transformed to the Reference Range according to the formula below.
- b) For reporting and analyzing, the data for females are linearly transformed to the Reference Range

- for males according to the formula below.
- c) For reporting and analyzing, the data are linearly transformed to the Reference Range according to the formula below.
  - To prevent transformed values becoming negative, the investigator lower limit is replaced by zero.
- d) Note that baseline values of 5 and 6 do not allow a subsequent clinically relevant change.
- e) To be done if dipstick is positive and microscopic examination needed for specific quantitation/confirmation.
- f) Specific gravity is a measurement of solute load in the urine. It is increased markedly by both proteinuria and glycosuria.

A value > 1.030 in the absence of proteinuria or glycosuria is most commonly caused by radiographic contrast. In volume depletion specific gravity is usually >1.020. A fixed value of 1.010 (isosthenuria) is characteristic of chronic renal impairment. A fixed value of 1.000 - 1.005 occurs in diabetes insipidus. Specific gravity has an important influence on urine microscopy because cells lyse more rapidly in dilute urine, which may lead to considerable inaccuracies in quantitation of cells. Cells swell and rupture in dilute urine and shrink in concentrate urine. Casts are rarely seen at low urine osmolality [5].

Conclusion: increase or decrease in urine specific gravity clinically relevant in context with other parameters from urinalysis.

Note: The following modification is applied to creatinine and TSH as needed.

Creatinine: The transformation of data described above as c) is applied for only Japanese patients study as needed.

TSH: The lower limit of the reference range and Marked Abnormal Range are modified and Clinically Relevant Change from Baseline for decrease is provided as needed.

• Formula for Linear Transformation

$$R_T = S_L + [(R_U - I_L) / (I_H - I_L)]*(S_H - S_L)$$

R<sub>T</sub>: transformed value

R<sub>U</sub>: untransformed value

Related to: SOP-GDO-WW-019

I<sub>L</sub>: IH investigator limits, low and high

S<sub>L</sub>: SH reference limits, low and high

For female to male transformation replace  $I_L$ ,  $I_H$  by the reference limits for female, and  $S_L$ ,  $S_H$  by the reference limits for male.

## 7.6 Rule for summary of titer for anti AQP4 antibody status

Titer for anti AQP4 antibody status except screening visit will be replaced by following rule. This rule will apply to throughout TFL.

- If value is "<16", value will be replaced as 4.
- If titer is character (e.g. ">16384", ">65536" except "<16") or titer is numeric more than 16384 (e.g. "65536", "262144"), value will be replaced as 65536.

